# University of California, San Francisco Clinical Research Protocol

# The TLC Study: Treatment with Lorcaserin for Cocaine Use

| Protocol Number: | 17-21502 |
|--------------------------|-------------------------------------------|
| Version Date: | 7/22/2017 |
| Investigational Product: | BELVIQ® XR (lorcaserin) |
| IND Number: | 134951 |
| Development Phase: | Phase II |
| Sponsor: | Glenn-Milo Santos, PhD, MPH |
| | University of California at San Francisco |
| | Department of Community Health Systems |
| | School of Nursing |
| | 2 Koret Way, N505 |
| | San Francisco, California 94143-0608 |
| Funding Organization: | National Institute on Drug Abuse (NIDA) |
| Principal Investigator: | Name: Glenn-Milo Santos, PhD, MPH |
| | Telephone: (628) 217-6231 |
| | E-mail: Glenn-milo.Santos@ucsf.edu |
| Medical Monitor: | Name: Phillip Coffin, |
| | Telephone: (510) 407-2603 |
| | E-mail: Phillip.coffin@sfdph.org |
| Coordinating Center: | San Francisco Department of Public Health |
| | Population Health Division |
| | 25 Van Ness Avenue, Suite 500 |
| | San Francisco, California 94102 |

| Approval: | |
|------------------------------------------|------------|
| Jan Jah | 07-22-2017 |
| PI or Sponsor Signature (Name and Title) | Date |

This confidential information about an investigational product is provided for the exclusive use of investigators of this product and is subject to recall at any time. The information in this document may not be disclosed unless federal or state law or regulations require such disclosure. Subject to the foregoing, this information may be disclosed only to those persons involved in the study who have a need to know, with the obligation not to further disseminate this information.

Version 2: Version Date: 7/22/2017 

# PROTOCOL AGREEMENT

I have read the protocol specified below. In my formal capacity as Investigator, my duties include ensuring the safety of the study subjects enrolled under my supervision as outlined in the protocol. It is understood that all information pertaining to the study will be held strictly confidential and that this confidentiality requirement applies to all study staff at this site. Furthermore, on behalf of the study staff and myself, I agree to maintain the procedures required to carry out the study in accordance with accepted GCP principles and to abide by the terms of this protocol.

| Protocol Number | r: 17-21502 | |
|---|---|---|
| Protocol Title: T | The TLC Study: Treatment with Lorcasering | for Cocaine Use |
| Protocol Date: T | TBD | |
| Janga | A | 07-22-2017 |
| Investigator Sign | nature | Date |
| Glenn-Milo Sant | os, Associate Professor | |
| Print Name and | Title | |
| Site # | 1 | |
| Site Name | San Francisco Department of Public Health | |
| Address | 25 Van Ness Ave, Suite # 500 | |
| | San Francisco, CA. 94102 | |
| Phone Number | | |

# TABLE OF CONTENTS

| 1 | BAC | CKGROUND1 | 10 |
|----|------|--------------------------------------------------|--------|
| | 1.1 | Overview of Clinical Studies | 0 |
| 2 | STU | DY RATIONALE1 | 12 |
| | 2.1 | Risk / Benefit Assessment | 2 |
| 3 | STU | DY OBJECTIVES1 | 13 |
| | 3.1 | Primary Objective1 | 13 |
| | 3.2 | Secondary Objectives | 13 |
| 4 | STU | DY DESIGN | 14 |
| | 4.1 | Study Overview | 4 |
| 5 | CRI | TERIA FOR EVALUATION1 | 14 |
| | 5.1 | Primary Efficacy Endpoint | 4 |
| | 5.2 | Secondary Efficacy Endpoints | 4 |
| | 5.3 | Safety Evaluations | Error! |
| | | kmark not defined. | |
| 6 | SUB | JECT SELECTION1 | |
| | 6.1 | Study Population1 | |
| | 6.2 | Inclusion Criteria | 4 |
| | 6.3 | Exclusion Criteria | 15 |
| 7 | CON | NCURRENT MEDICATIONS1 | 15 |
| | 7.1 | Allowed1 | 15 |
| | 7.2 | Prohibited1 | 15 |
| 8 | STU | DY TREATMENTS | 15 |
| | 8.1 | Method of Assigning Subjects to Treatment Groups | 15 |
| | 8.2 | Blinding1 | 16 |
| | 8.3 | Test and Control Formulation | 16 |
| | 8.4 | Supply of Study Medication at the Site | Error! |
| | | kmark not defined. | |
| | 8.5 | Study Medication Accountability | |
| _ | 8.6 | Measures of Treatment Compliance 1 | |
| 9 | | DY PROCEDURES AND GUIDELINES1 | |
| | 9.1 | Clinical Assessments | |
| | 9.2 | Clinical Laboratory Measurements | |
| 10 | | ALUATIONS BY VISIT2 | |
| | | Visit 1 (Screening 1 Visit) | |
| | | Visit 2 (Screening 2 Visit) | |
| | | Visit 3 (Enrollment) | |
| | | Visit 4 (Weekly Visits) | |
| | | Visit 5 (Monthly) | |
| | 10.6 | Early Withdrawal Visit | 23 |

| 11 | ADV | ERSE EXPERIENCE REPORTING AND DOCUMENTATION | 23 |
|---|---|---|---|
| | 11.1 | Adverse Events | 23 |
| | 11.2 | Serious Adverse Experiences (SAE) | 25 |
| | 11.3 | Protocol Defined Important Medical Findings Requiring Real Time Reporting | Error! |
| | Book | kmark not defined. | |
| | | Medical Monitoring | Error! |
| | | kmark not defined. | |
| | | Safety Management Plan | |
| | | CONTINUATION AND REPLACEMENT OF SUBJECTS | ERROR! |
| BO | | ARK NOT DEFINED. | Б. |
| | | Withdrawal of Subjects | Error! |
| | | Replacement of Subjects | Errort |
| | | kmark not defined. | Effor: |
| 13 | | TOCOL VIOLATIONS | ERROR! |
| | | ARK NOT DEFINED. | Litatoit. |
| 14 | DAT | A SAFETY MONITORING | ERROR! |
| ВО | OKM | ARK NOT DEFINED. | |
| _ | | TISTICAL METHODS AND CONSIDERATIONS | ERROR! |
| ВО | | ARK NOT DEFINED. | |
| | | Data Sets Analyzed | Error! |
| | | kmark not defined. | |
| | | Demographic and Baseline Characteristics | Error! |
| | | | 20 |
| | | Analysis of Primary Endpoint | |
| | | Analysis of Secondary Endpoints | |
| | | Interim Analysis | |
| 1. | | Sample Size and Randomization | |
| 16 | | A COLLECTION, RETENTION AND MONITORING | |
| | | Data Collection Instruments | |
| | | Data Management Procedures | |
| | | Data Quality Control and Reporting. | |
| | | Archival of Data | |
| | | Availability and Retention of Investigational Records | |
| | | Monitoring | |
| | | Subject Confidentiality | |
| 17 | | IINISTRATIVE, ETHICAL, REGULATORY CONSIDERATIONS | |
| | | Protocol Amendments | |
| | 17.2 | Institutional Review Boards and Independent Ethics Committees | |
| | 17.3 | Informed Consent Form | |
| | | Publications | |
| | | Investigator Responsibilities | |
| 18 | APPI | ENDICES | 36 |

| PI: Santos, Glenn-Milo | Confidential |
|------------------------|--------------|

| 18.1 | Study Procedures | 36 |
|------|------------------|----|
| 18.2 | References | 36 |

#### LIST OF ABBREVIATIONS

ACASI Audio Computer Assisted Survey Instrument

**AE** adverse event

ALT alanine aminotransferase
AST aspartate aminotransferase

**BART** Balloon Analogue Risk Task – impulsivity test

BMI Body Mass Index
BUN blood urea nitrogen
CBC Complete blood count

CBO Community based organization
CCG Community Consulting Group
CFR Code of Federal Regulations

**CRF** case report form

CPHR Center for public health research

DMC Data Monitoring Committee

DSMB Data Safety Monitoring Board

**DSM-IV** Diagnostic and Statistical Manual for Mental disorders

**FDA** Food and Drug Administration

**GCP** Good Clinical Practice

**GEE** generalized estimating equations

HIPAA Health Insurance Portability and Accountability Act of 1996

HIV Human Immunodeficiency Virus

**ICF** informed consent form

ICH International Conference on Harmonisation

IEC Independent Ethics Committee
IRB Institutional Review Board

MM Medical Management counseling
MSM Men who have sex with men

NIAAA National Institute on Alcohol Abuse and Alcoholism

PrEP pre-exposure prophylaxis
PI Principal Investigator
SAE serious adverse experience

**SAMHSA** Substance Abuse and Mental Health Services Administration

SCID Structural clinical interview for DSM disorders
SFDPH San Francisco Department of Public Health

SMS Text message

**TLFB** Timeline follow-back

# PROTOCOL SYNOPSIS

| TITLE | The TLC Study: Treatment with Lorcaserin for Cocaine Use |
|---|---|
| SPONSOR | Glenn-Milo Santos |
| FUNDING<br>ORGANIZATION | NIDA |
| NUMBER OF SITES | 1 |
| RATIONALE | Lorcaserin's mechanism of action as a potent 5-HT <sub>2C</sub> R selective agonist may have inhibitory control on DA activity, which may decrease the positive rewarding effects of cocaine and lead to reductions in use, while 5-HT <sub>2C</sub> R activation itself may lead to reductions in likelihood of relapse. There are no pharmacological agents available to reduce cocaine use disorder. |
| STUDY DESIGN | This study will enroll 45 actively using Men who have sex with men with cocaine use disorders in a placebo-controlled 12-week trial. Individuals will be randomly assigned (2:1) to receive 12 weeks of lorcaserin 20mg (n=30) or placebo (n=15) to be taken daily in this double-blind trial. |
| PRIMARY<br>OBJECTIVE | To establish the feasibility, tolerability, acceptability and adherence of enrolling and retaining 45 adults with cocaine use disorders in a 12-week randomized, double-blind study of lorcaserin versus placebo. |
| SECONDARY<br>OBJECTIVES | To evaluate the <u>preliminary efficacy</u> of lorcaserin versus placebo to reduce cocaine use and HIV-related sexual risk behaviors among MSM with cocaine use disorders, as determined by the proportion of cocaine-positivity from twice weekly urine samples and self-reported sexual behaviors. |
| NUMBER OF<br>SUBJECTS | 45 |
| SUBJECT<br>SELECTION<br>Criteria | Inclusion Criteria: 1) Male gender; 2) self-reported anal intercourse with men in the prior six months while under the influence of cocaine; 3) cocaine use disorder by DSM-V SCID criteria; 4) current cocaine use confirmed by urinalysis and cocaine use at least 1 day in the past 30 days; 5) HIV-negative by rapid test or HIV-positive with medical record of HIV infection; 6) no current acute illnesses requiring prolonged medical care; 7) no chronic illnesses that are likely to progress clinically during trial; 8) able and willing to provide informed consent and adhere to visit schedule; 9) age 18–65 years; 10) baseline CBC, total protein, albumin, glucose, alkaline phosphatase, creatinine, BUN, and electrolytes without clinically significant abnormalities as determined by study clinician in conjunction with symptoms, physical exam, and medical history. |
| | Exclusion Criteria: 1) Any psychiatric condition (e.g., depression with suicidal ideation, schizophrenia) or medical condition that would preclude safe study participation; 2) HIV-positive test result at screening visit but previously unaware of HIV infection (i.e., newly diagnosed with HIV infection at screening; those with a medical record of HIV infection are |


| | eligible); 3) any moderate to severe alcohol or substance use disorders (other than cocaine use disorders), according to DSM-V criteria; 4) known allergy or previous adverse reaction to lorcaserin; 5) current CD4 count < 200 cells/mm3; 6) severe liver impairment (Child-Pugh score > 9); 7) severely impaired renal function (creatinine clearance £ 30 ml/min); 8) use of medications that affect the serotonergic neurotransmitter system (e.g., selective serotonin reuptake inhibitors (SSRIs), selective serotoninnorepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, monoamine oxidase inhibitors (MAOIs)); 9) predisposition to priapism; 10) currently participating in another longitudinal intervention research study; 11) body mass index (BMI) $\geq$ 30 with desire to use weight management medication, or BMI > 40;12) BMI < 15; 13) anticipated use of agents that are associated with valvulopathy and/or pulmonary hypertension |
|---|---|
| TEST PRODUCT, DOSE, AND ROUTE OF ADMINISTRATION | BELVIQ® XR (lorcaserin) 20mg., manufactured by: Arena Pharmaceuticals: Untere Brühlstrasse 4, 4800 Zofingen, Switzerland Product will be administered orally each day for 12 weeks length of time. |
| CONTROL PRODUCT, DOSE AND ROUTE OF ADMINISTRATION | Placebo, 20 mg. Product will be administered orally each day for 12 weeks length of time. |
| DURATION OF<br>SUBJECT<br>PARTICIPATION<br>AND DURATION OF<br>STUDY | Subjects will be on study for up to 12 weeks Screening: up to 4 weeks Treatment: 12 weeks The total duration of the study is expected to be 16 weeks or 4 months. 1 month for subject recruitment and 3 months for treatment phase. |
| CONCOMMITANT<br>MEDICATIONS | Allowed: standard treatment Prohibited: Serotonin reuptake inhibitors (SSRIs), selective serotonin- norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, monoamine oxidase inhibitors (MAOIs) |
| EFFICACY<br>EVALUATIONS | |
| PRIMARY ENDPOINT | In the overall sample of 45, proportions will be estimated with margins of sampling error (MSEs; i.e., half widths of 95% confidence intervals) of <=14.4 percentage points, and means with MSEs of 0.30 standard deviations, both typical for a small pilot study. While the study will only be powered to detect large between-group differences in process measures, it will provide warning of potential problems. |
| SECONDARY<br>ENDPOINTS | We will also classify AEs as any AE that results in stopping study medication, specific common AEs (>2% in both groups), AEs for general |


| | organ system categories, and AEs potentially related to study drug. The probability of observing at least one AE with population incidence of 1, 2, and 5% in the active arm will be 26, 45, and 70% with 2:1 randomization, respectively. |
|---|---|
| SAFETY<br>EVALUATIONS | Change in clinical safety labs from baseline to Week 12 Incidence of adverse events |
| PLANNED INTERIM<br>ANALYSES | No planned interim analyses |
| STATISTICS Primary Analysis Plan | To establish the feasibility of enrolling and retaining 45 MSM with cocaine use disorders in a 12-week 2:1 randomized, double-blind study of lorcaserin versus placebo. We will calculate the following feasibility measures: 1) proportion of those eligible among those screened; 2) proportion enrolled among those eligible; and 3) study completion rate. Process measures (e.g., visit length, counseling session completion) and reactions to study procedures will also be collected and reported. Between-group differences will be assessed using Fisher's exact and Wilcoxon rank sum tests. We will also calculate Kaplan-Meier curves for time to dropout, by group, and test for differences using the log-rank test. Precision: In the overall sample of 45, proportions will be estimated with margins of sampling error (MSEs; i.e., half widths of 95% confidence intervals) of ≤14.4 percentage points, and means with MSEs of 0.30 standard deviations, both typical for a small pilot study. While the study will only be powered to detect large between-group differences in process measures, it will provide warning of potential problems. To explore the tolerability of lorcaserin versus placebo among MSM with cocaine use disorders, as determined by the number of adverse clinical events in the cocaine and placebo arms. We will compute the proportions of those experiencing adverse events, both overall and by type. Adverse clinical events, AEs and SAEs, and other binary safety outcomes will be presented as percent of participants that experience the safety outcome by treatment assignment. We will also classify AEs as any AE that results in stopping study medication, specific common AEs (>2% in both groups), AEs for general organ system categories, and AEs potentially related to study drug. The probability of observing at least one AE with population incidence of 1, 2, and 5% in the active arm will be 26, 45, and 70% with 2:1 randomization, respectively. To describe the acceptability and adherence for lorcaserin versus placebo MSM with cocaine |


| Rationale for Number of Subjects | In the overall sample of 45, proportions will be estimated with margins of sampling error (MSEs; i.e., half widths of 95% confidence intervals) of ≤14.4 percentage points, and means with MSEs of 0.30 standard deviations, both typical for a small pilot study. While the study will only be powered to detect large between-group differences in process measures, it will provide warning of potential problems. |
|---|---|

# 1. BACKGROUND

Lorcaserin, a novel selective serotonin (5-HT) receptor agonist, is a promising agent to treat cocaine use disorders. Cocaine use increases dopamine (DA) levels, the neurochemical responsible for the reinforcing effects of the drug, and there is compelling data suggesting that the DA system's activity is modulated by the central 5-HT systems.<sup>69-71</sup>

In particular, the 5-HT<sub>2C</sub> receptor (5-HT<sub>2C</sub>R) has been identified as the primary 5-HT receptor subtype that inhibits the DA system's activity.  $^{71}$  5-HT<sub>2C</sub>R agonists have reduced dopamine release in the nucleus accumbens (NAcc) and frontal neurocortex. 69,71 Conversely, increased DA release in the NAcc result from the blockade of 5-HT<sub>2C</sub>R.  $^{72}$ 

#### **OVERVIEW OF CLINICAL STUDIES**

Cocaine use in the US is an *unrelenting public health problem* with serious negative medical, societal, and economic impacts. <sup>1-3</sup> The US is the world's largest consumer of cocaine, accounting for nearly

36% of the total global consumption. <sup>4,5</sup> In both powder and rock (i.e., "crack") form, cocaine is an addictive psychostimulant; it is estimated that up to one in six cocaine users may develop dependence/moderate-to-severe use disorders. Cocaine is the leading cause of illicit substance–related emergency department visits in the US and it is associated with direct cardiac toxicity, myocardial infarctions and, sudden cardiac death. Cocaine use is a significant decrease (test for trend p<0.001) <sup>17,18</sup> in



methamphetamine use among San Francisco MSM (from 22% to 13%). San Francisco communitybased surveys observed similar trends: cocaine use among MSM increased from 9.6% in 2009 to 20.4% in 2013. 19,20 Of the estimated 19,657 illicit psychostimulant- using MSM in San Francisco, 81.3% are cocaine users. 16 MSM remain disproportionately impacted by HIV—despite sizable efforts to stem the epidemic in this group—accounting for 61% and 90% of new infections in the US and San Francisco, respectively. 21-24 It is imperative to develop more evidence-based HIV interventions for MSM; the National HIV/AIDS Strategy specifically calls for additional interventions for this population. <sup>25</sup> Cocaine use is associated with HIV-related sexual risk behaviors in MSM. In NHBS, 54% of cocaine users reported having sex while under the influence of cocaine. <sup>14</sup> The acute pharmacological effects of cocaine (e.g., altered cognition, impairment of judgment, and increased sexual desire and confidence) have been attributed to the association between cocaine use and sexual risk behaviors. 26-30 Moreover, a myriad of psychosocial factors (e.g., cognitive escape, impulsivity, and expectancies) are thought to account for the link between cocaine use and sexual risks. 31-34 Furthermore, the bar, club, and circuit-party (weekend-long dance events) settings frequented by MSM are environments conducive to both cocaine use and meeting multiple sex partners. 35-37 Indeed, cocaine use is independently associated with unprotected anal intercourse, multiple partners, increased duration of sex, anonymous partners, sex in a public sex venue, and exchanging money or drugs for sex. 38-43 In the Project ECHO study, a large San Francisco study of substance-using MSM conducted by the proposed research team, increased frequency of cocaine use was associated with greater HIV-related sexual risk; those who reported episodic use (less than weekly) and those with weekly or greater cocaine use had 1.86- and 3.13-fold greater odds of HIV serodiscordant unprotected anal intercourse,

respectively, compared to non-users. <sup>44</sup> This dose-dependent relationship is consistent with findings from a probability sample of HIV-negative MSM; those with cocaine dependence were more likely to have high-risk sexual behaviors than their non-dependent counterparts. <sup>41</sup>

Cocaine use has been significantly associated with new HIV infections. 45-47 In the EXPLORE longitudinal study of 4,295 HIV-negative MSM from six cities, cocaine use was associated with a 2.24-fold greater hazard for HIV seroconversion. Similarly, in the Multicenter AIDS Cohort Study, use of cocaine or other stimulants, alone or in combination with other drugs, was attributed to 37.3% of the new HIV infections in the study. In a probability sample of San Francisco MSM, cocaine and other stimulant use was also 2.5-fold more common among MSM living with HIV. Among HIV-positive individuals, cocaine use was associated with poor adherence to antiretroviral treatment (ART), HIV disease progression, lower CD4 count, and higher mortality. Weekly cocaine use was associated with higher HIV viral load, even after controlling for ART adherence, and in *in vitro* studies, cocaine enhanced HIV viral replication. Poor ART adherence and higher HIV viral load among cocaine users may potentiate greater risk of HIV transmission.

Innovative treatments for cocaine use disorders are needed for MSM. 57 Because cocaine use is common among MSM and is associated with high-risk sexual behavior and HIV infection, interventions that can reduce cocaine use are likely to have an impact on reducing the transmission of HIV. 28 Current prevention approaches to cocaine use for MSM are therapy and substance use treatment programs. However, most substance-using MSM do not access drug treatment, reinforcing the need to develop interventions outside of treatment settings. 44,58,59 Furthermore, while some behavioral interventions for substance-using MSM report reductions in both substance use and HIV risk  $behaviors, ^{60,61} behavioral\ interventions\ alone\ have\ limited\ efficacy\ and\ may\ benefit\ from\ adjuvant$ pharmacologic agents However, there are no FDA-approved medications for cocaine use disorders, which severely limits treatment options. <sup>63,64</sup> Pharmacologic approaches have been successful in treating nicotine, alcohol, and heroin dependence. Despite the link between cocaine use and HIV risk, the use of pharmacologic interventions to reduce cocaine-related sexual risk among MSM remains underexplored. The absence of published studies on efficacious interventions to reduce cocaine- related sexual risk behaviors among MSM who have no desire to abstain from cocaine presents a major gap in the field of substance use research and HIV prevention. Pharmacotherapy for methamphetamine dependence in MSM has shown that reductions in substance use can result in parallel reductions in methamphetamine-related sexual risk behaviors among MSM not seeking treatment. 68 Pharmacotherapy for cocaine use may lead to an analogous parallel reduction in cocainerelated sexual risks.

**Lorcaserin, a novel selective serotonin (5-HT) receptor agonist, is a promising agent to treat cocaine use disorders.** Cocaine use increases dopamine (DA) levels, the neurochemical responsible for the reinforcing effects of the drug, and there is compelling data suggesting that the DA system's activity is modulated by the central 5-HT systems.<sup>69-71</sup> In particular, the 5-HT<sub>2C</sub> receptor (5-HT<sub>2C</sub>R) has been identified as the primary 5-HT receptor subtype that inhibits the DA system's activity.<sup>71</sup> 5-HT<sub>2C</sub>R agonists have reduced dopamine release in the nucleus accumbens (NAcc) and frontal neurocortex. Conversely, increased DA release in the NAcc result from the blockade of 5-HT<sub>2C</sub>R.<sup>72</sup> Furthermore,


genetic variations in the 5-HT<sub>2C</sub>R and its functional status have been associated with vulnerability to cocaine cue reactivity—a strong predictor of relapse—and relapse- like behaviors in cocaine dependent rodents and humans. These data lend support to the use of agents that selectively activate the 5- $HT_{2C}R$ . We postulate that lorcaserin's mechanism of action as a potent 5-HT<sub>2C</sub>R selective agonist will have inhibitory control on DA activity, which may decrease the positive rewarding effects of cocaine and lead to reductions in use, while 5-HT<sub>2C</sub>R activation itself may lead to reductions in likelihood of relapse.

Preclinical data support the potential of lorcaserin in reducing cocaine use. To,75-85 Lorcaserin is 18- and 120-fold more selective toward the 5-HT<sub>2C</sub>R compared to 5-HT<sub>2A</sub> and 5-HT<sub>2B</sub> receptors, respectively. Lorcaserin is 18- and 5-HT<sub>2C</sub>R selective agonists, including lorcaserin, have been associated with reductions in cocaine self-administration in mice and non-human primates. Consistent reductions in cue- and cocaine-primed drug seeking have resulted from use of 5-HT<sub>2C</sub>R selective agonists. Furthermore, 5-HT<sub>2C</sub>R selective agonists have attenuated acute cocaine-induced activity and the development of long-term cocaine-induced locomotor sensitization. Reinstatement studies to model the relapse processes have also found that 5-HT<sub>2C</sub>R selective agonists reduced cocaine seeking behavior, again in both rodents and primates.

Data from other preclinical and clinical studies also support lorcaserin's potential to treat drug disorders. For example, lorcaserin has been shown to reduce nicotine self-administration, <sup>95</sup> as well as nicotine discrimination, and cue-induced reinstatement of nicotine seeking. <sup>96</sup> Currently, another team is evaluating lorcaserin in a placebo-controlled Phase 2, 12-week trial on smoking cessation (ClinicalTrials.gov #: NCT02044874).

#### 2. STUDY RATIONALE

## 2.1 Study Overview:

This study will represent the *first* Phase 2 randomized outpatient clinical trial to evaluate the potential of lorcaserin to reduce cocaine use among actively using participants with cocaine use disorders. Although there is an ongoing human laboratory study of lorcaserin's effects on craving and intravenous cocaine self-administration during overnight confinements at a medical center (ClinicalTrials.gov #: NCT02680288), our proposed study will provide distinct yet complementary data on the viability of lorcaserin to reduce cocaine. Our study is unique because it involves the outpatient treatment and evaluation of lorcaserin to reduce cocaine use and cocaine-associated sexual risk behaviors among men who have sex with men *over a 12-week follow-up period*. Hence, data from this pilot can inform the sample size required for a larger clinical efficacy trial of lorcaserin for outpatient treatment of cocaine use. Additionally, this study will determine if lorcaserin is a feasible, tolerable, and acceptable option for cocaine outpatient treatment.

#### 2.2 Risk / Benefit Assessment

**Lorcaserin is an FDA-approved medication that is well-tolerated with relatively few adverse events (AEs).** Three Phase 3 trials (cumulative N=7789) that evaluated lorcaserin's treatment effect on obesity have established its safety among patients with and without diabetes. The most


common reported side effects for lorcaserin include headaches, dizziness, fatigue, nausea, dry mouth, and constipation. In these trials, 8.6% of individuals given lorcaserin discontinued treatment as a result of AEs, compared to 6.7% individuals given placebo. Aside from pregnancy, there are no contraindications for lorcaserin. Nevertheless, the safety and tolerability of lorcaserin among active cocaine users is unknown. Lorcaserin has a low potential for abuse. The frequency of AEs associated with lorcaserin increases when taken above the therapeutic dose, which may limit abuse potential. A double-blind randomized crossover study to test abuse liability found that lorcaserin was similar to placebo with respect to subjective liking, overall liking, and ratings on desire to take the drug again. Exceeding the recommended lorcaserin dose levels (10 mg, twice daily) were associated with higher levels of known unpleasant side effects and subjective dislike, compared to placebo. Thus, lorcaserin dose escalation would result in primarily negative subjective effects; these self-regulating properties will likely limit the medication's abuse liability.

#### 3. STUDY OBJECTIVES

# 3.1 Primary Objective

The primary objective is to evaluate the feasibility, tolerability, acceptability and adherence of lorcaserin versus placebo (2:1) to reduce cocaine use disorder among 45 MSM cocaine users over 12 week treatment period.

# 3.2 Secondary Objectives

To evaluate the <u>preliminary efficacy</u> of lorcaserin versus placebo to reduce cocaine use and HIV-related sexual risk behaviors among MSM with cocaine use disorders, as determined by the proportion of cocaine-positivity from twice weekly urine samples and self-reported sexual behaviors over a 12 week treatment period.

#### 4. STUDY DESIGN

## 4.1 Study Overview

The goal of the TLC Study is to evaluate the *feasibility, tolerability, acceptability* and *adherence* for lorcaserin among actively using, MSM with cocaine use disorders in a placebo-controlled 12-week trial. In a double-blind trial, 45 individuals will be randomly assigned (2:1) to receive 12 weeks of lorcaserin 20mg (n=30) or placebo (n=15), to be taken once a day.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

The following treatment regimens will be used:

- Experimental treatment: BELVIQ® XR (lorcaserin). 20 mg.
- Placebo or Comparator Placebo, 20 mg.


Total duration of subject participation will be twelve weeks. Total duration of the study is expected to be 16 weeks.

#### 5. CRITERIA FOR EVALUATION

# 5.1 Primary Efficacy Endpoint

For the primary efficacy endpoint, we conservatively estimate that the sample will provide 80% power to detect reductions of 29 percentage points in the rate of cocaine urine positivity. The time course for which this endpoint will be assessed will be from baseline to 12 week end of treatment. We will also evaluate between-group differences on changes in: 1) any cocaine positive samples, defined as having a positive urine or sweat patch sample, over follow-up; 2) any cocaine positive samples or self-report of cocaine use in text messages; and 3) cocaine positivity from sweat samples only.

# 5.2 Secondary Efficacy Endpoints

For the secondary efficacy endpoint, to evaluate treatment effects on cocaine-associated sexual risk behaviors, GEE Poisson, binomial, and negative binomial models will be used to assess treatment effects on HIV sexual risk behaviors including high-risk sexual behaviors while under the influence of cocaine.

# **5.3 Safety Evaluation:**

- Change in clinical laboratory findings
- Incidence of adverse events

#### 6. SUBJECT SELECTION

#### **6.1 Study Population**

Men who have sex with men with a diagnosis of cocaine use disorder who meet the inclusion and exclusion criteria will be eligible for participation in this study.

#### **6.2 Inclusion Criteria**

- 1) Male gender;
- 2) self-reported anal intercourse with men in the prior six months while under the influence of cocaine;
- 3) cocaine use disorder by DSM-V SCID criteria;
- 4) current cocaine use confirmed by urinalysis and cocaine use at least 1 day in the past 30 days;
- 5) HIV-negative by rapid test or HIV-positive with medical record of HIV infection;
- 6) no current acute illnesses requiring prolonged medical care;
- 7) no chronic illnesses that are likely to progress clinically during trial;
- 8) able and willing to provide informed consent and adhere to visit schedule;
- 9) age 18–65 years;
- 10) Baseline CBC, total protein, albumin, glucose, alkaline phosphatase, creatinine, BUN, and electrolytes without clinically significant abnormalities as determined by study clinician in conjunction with symptoms, physical exam, and medical history.
- 11) Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.


#### 6.3 Exclusion Criteria

1) Any psychiatric condition (e.g., depression with suicidal ideation, schizophrenia) or medical condition that would preclude safe study participation;

- 2) HIV-positive test result at screening visit but previously unaware of HIV infection (i.e., newly diagnosed with HIV infection at screening; those with a medical record of HIV infection are eligible);
- 3) any moderate to severe alcohol or substance use disorders (other than cocaine use disorders), according to DSM-V criteria;
- 4) known allergy or previous adverse reaction to lorcaserin;
- 5) current CD4 count < 200 cells/mm3;
- 6) severe liver impairment (Child-Pugh score > 9);
- 7) severely impaired renal function (creatinine clearance £ 30 ml/min);
- 8) use of medications that affect the serotonergic neurotransmitter system (e.g., selective serotonin reuptake inhibitors (SSRIs), selective serotonin- norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, monoamine oxidase inhibitors (MAOIs));
- 9) predisposition to priapism;
- 10) currently participating in another longitudinal intervention research study;
- 11) body mass index (BMI)  $\geq$  30 with desire to use weight management medication, or BMI > 40;
- 12) BMI < 15; 13) anticipated use of agents that are associated with valvulopathy and/or pulmonary hypertension

#### 7. CONCURRENT MEDICATIONS

All subjects should be maintained on the same medications throughout the entire study period, as medically feasible, with no introduction of new chronic therapies.

### 7.1 Allowed Medications and Treatments

Standard therapy is allowed except for treatments noted in the exclusion criteria described above and as noted in the prohibited medications section below.

## 7.2 Prohibited Medication and Treatments

No prohibited medication or treatment besides those in the exclusion criteria.

#### 8. STUDY TREATMENTS

# 8.1 Method of Assigning Subjects to Treatment Groups

Up to 45 eligible participants will be randomly assigned to lorcaserin or placebo treatment groups in a 2:1 allocation ratio (lorcaserin and placebo), using the computer-generated randomization code for the study blocks. Assignment of two-thirds of participants to the lorcaserin arm was specifically chosen to improve our ability to detect adverse events in the active treatment arm, while preserving our ability to assess recruitment in a study in which randomization to placebo is likely. The study biostatistician, Dr.


Vittinghoff, will generate and provide the randomization code directly to the pharmacy. No study staff will have access to the code.

# 8.2 Blinding

Due to the objectives of the study, the identity of test and control treatments will not be known to investigators, research staff, or participant. The following study procedures will be in place to ensure double-blind administration of study treatments.

Access to the randomization code will be strictly controlled.

Packaging and labeling of test and control treatments will be identical to maintain the blind.

The study blind will be broken on completion of the clinical study and after the study database has been locked.

During the study, the blind may be broken **only** in emergencies when knowledge of the patient's treatment group is necessary for further patient management. When possible, the Investigator should discuss the emergency with the Medical Director prior to unblinding.

#### 8.3 Formulation of Test and Control Products

Drug Name and Active Ingredients

Name(s): BELVIQ® XR

Active Ingredients: lorcaserin hydrochloride

Pharmacological Class

BELVIQ® XR (lorcaserin hydrochloride) is a serotonin 2C receptor agonist for oral administration used for chronic weight management. [1]

Structural and Chemical Formula

Its chemical name is (R)-8-chloro-1-methyl-2,3,4,5-tetrahydro-1H-3-benzazepine hydrochloride hemihydrate. The empirical formula is C H Cl N·0.5H O, and the molecular weight of the hemihydrate form is 241.16 g/mol.[1]

The structural formula is:

Formulation of Dosage

This drug is in the form of an orange, film-coated, round, film-coated, 20 mg extended release tablet. The tablets are biconvex, debossed with "A" on one side and "20" on the other side

For this investigation, BELVIQ® XR will not be compounded. We will have Safeway Pharmacy (located at 6100 Hellyer Avenue, Suite 100 San Jose, CA 95138) encapsulate the BELVIQ® XR pill in whole form and create identical placebo capsules.[1]

Route of Administration

#### **Packaging and Labeling**

Safeway Compounding Pharmacy, 6100 Hellyer Ave Ste 100, San Jose, CA, 95138, is used to provide study drug. Each treatment bottle from the UCSF pharmacy was labeled with the study drug number, prescribing physician name (medical director), required FDA warning statement, emergency pager number, directions for participant use and storage, and expiration information. Each treatment bottle from Safeway pharmacy is labeled with the study drug number, principal investigator name, prescribing physician name (medical director), required FDA warning statement, emergency pager number, directions for participant use and storage, and lot and expiration information.

#### Sample Label:



# 8.4 Supply of Study Drug at the Site

The Safeway Compounding Pharmacy (San Jose, CA), which is currently supplying the study drug for our ongoing trials, will prepare and supply lorcaserin and placebo in identical-looking gel capsules to maintain blinding. The initial study drug shipment will be shipped after site activation (i.e., all required regulatory documentation has been completed). Subsequent study drug shipments will be made after site request for resupply.

# 8.4.1Dosage/Dosage Regimen

The recommended dose of BELVIQ® XR is one 20mg tablet administered orally once daily.[1]

#### 8.4.2 Dispensing

Study medications will be dispensed by the study clinician (licensed medical practitioner) in treatment bottles that are labeled with the study drug number, principal investigator name, prescribing physician name (medical director), required FDA warning statement, emergency pager number, directions for participant use and storage, and lot and expiration information.

Further, at time of study drug dispensing, the study clinician will review with the participant how to take the study medication, possible side effects they may encounter, and how to access the study clinician by emergency pager if necessary. The study clinician will also answer any questions the participant might have.

#### **8.4.3** Administration Instructions

Participants will receive training on dosing at enrollment. Participants will be given a week's supply of 20mg tablets at enrollment and at weekly visits; they will be instructed to only take 1 tablet every 24 hours. This optimal dose was informed by pharmacokinetic studies which estimated that 20mg of lorcaserin has a mean plasma half-life of 11 hours and once daily 20mg dosing of lorcaserin will lead to steady state within 3 days of treatment. <sup>104</sup>

## 8.4.4 Storage

Study drug should be stored by the study site at controlled room temperature, 15 to 30°C (59 to 86°F). If the temperature of study drug storage in the clinic/pharmacy exceeds or falls below this range, this should be reported to the Principal Investigator and captured as a deviation. Subjects will be instructed to store the medication in original packaging at room temperature according to the instructions outlined on the Drug Administration Instructions.

## 8.5 Study Drug Accountability

An accurate and current accounting of the dispensing and return of study drug for each subject will be maintained on an ongoing basis by a member of the study site staff. The number of study drug dispensed and returned by the subject will be recorded on the Investigational Drug Accountability Record.

# 8.6 Measures of Treatment Compliance

Study medications will be dispensed by the study clinician in MEMs cap dispensers with dosing instructions, date of dispensing, prescribing clinician, a 24-hour telephone study phone number for medical emergencies, and advisements against drug combinations. MEMS Caps will track adherence daily; each dispenser opening is recorded as a medication event sent to a remote database in real time

#### 9. STUDY PROCEDURES AND GUIDELINES

A Schedule of Events representing the required testing procedures to be performed for the duration of the study is diagrammed in Appendix 1.

Prior to conducting any study-related activities, written informed consent and the Health Insurance Portability and Accountability Act (HIPAA) authorization must be signed and dated by the subject or subject's legal representative. If appropriate, assent must also be obtained prior to conducting any study-related activities.

#### 9.1 Clinical Assessments

#### **Concomitant Medications**

All concomitant medication and concurrent therapies will be documented at Baseline/Screening and at Month 1, Month 2 and Month 3 visits. Dose, route, unit frequency of administration, and indication for administration and dates of medication will be captured.

#### **Demographics**

Demographic information (date of birth, gender, race) will be recorded at Screening.

# **Balloon Analogue Risk Tast (BART)**

To better understand the mechanism in which lorcaserin may reduce cocaine and cocaine-associated sexual risk behaviors, we will evaluate lorcaserin's effect on impulsivity through two validated measures of impulsivity: the state impulsivity scale (the STIMP)<sup>183</sup> and the Balloon Analogue Risk Task (BART).<sup>182</sup> We will evaluate changes in cocaine craving by arm using the visual analog scale for craving<sup>187</sup> and the Minnesota cocaine craving scale.<sup>188</sup>

#### **Medical History**

Relevant medical history, including history of current disease, other pertinent respiratory history, and information regarding underlying diseases will be recorded at Screening.


# **Physical Examination**

A complete physical examination will be performed by the study clinician at Screening, Enrollment, Month 1, Month 2, and Month 3 visits. Qualified staff (MD, NP, RN, and PA) may complete the abbreviated physical exam at all other visits. New abnormal physical exam findings must be documented and will be followed by a physician or other qualified staff at the next scheduled visit.

# **Vital Signs**

Body temperature, blood pressure, pulse and respirations will be performed after resting for 5 minutes at Enrollment, Month 1, Month 2 and Month 3 visits

# **Electrocardiogram (ECG):**

The ECG will be administered during screening to assist in determination of participant eligibility and again at study exit (ie. week 12/Month 3) to assess safety at termination. The ECG tracings will be reviewed by a qualified medical clinician for accuracy at the site.

# Figure 6: PharmChekDrugs of Abuse Sweat Patch

ticinant **Bottom:** Used sweat

pouch and labeled before being shipped for testing (adapted from<sup>8</sup>).

# **Urinalysis for Cocaine Use**

Urinalysis for Cocaine Use: Urine samples will be collected once a week and tested for cocaine metabolites (benzoylecgonine) with EZ-SCREEN screening assays (MedTox Diagnostics, Inc., Burlington, NC). On average, cocaine is detectable in urine for approximately 72 hours. To detect use over weekends, when cocaine use is likely to be higher compared to the remainder of the week. Furthermore, the MedTox assays we will use for urine toxicology tests can also detect the following classes of substances: amphetamine, barbiturates, benzodiazepines, buprenorphine, methadone, methamphetamine, opiates, oxycodone, phencyclidine, propoxyphene and THC (cannabinoids).

# **Sweat Testing Using Perspiration Patches**

To further enhance our ability to detect cocaine use, we will also utilize tamper evident sweat patches—PharmChek Drugs of Abuse Sweat Patch (PharmChem, Inc., Fort Worth, Texas)—that absorb perspiration 24 hours per day, for up to 10 days of continuous wear. These patches will be tested for the presence of cocaine and cocaine metabolites, using testing procedures approved by the FDA since 1995. Pharmchek patch enzyme immunoassays to detect cocaine in sweat have been found to have 94-95% sensitivity and 91-99% specificity rates, compared to gas chromatography-mass spectrometry. At baseline visit, we will affix patches on all participants (see **Figure 6**). These patches have a semi-permeable membrane to allow oxygen, carbon dioxide and water vapor to pass through the patch, keeping the skin underneath sterile and healthy. At each weekly follow-up visit, we will replace the used patch worn since the prior visit and send those used patches for cocaine testing to PharmChem's laboratories. These patches will retain cocaine and cocaine

cocaine testing to PharmChem's laboratories. These patches will retain cocaine and cocaine metabolites for any use during the period it was worn. Hence, we anticipate no gaps in the window of detection for cocaine use. *Extra replacement patches* will be provided to participants at weekly visits, in anticipation of the rare event that a patch falls off prematurely; participants will be instructed to use a replacement patch when needed. Used patches will be collected and tested weekly. In sensitivity analyses, we will impute cocaine-positive results for weeks in which multiple patches were used or when patches fell off.

## **HIV Testing and Counseling:**

Participants will receive standard HIV risk reduction counseling <sup>168</sup> at screening and at month 3 visits with HIV rapid test and pooled viral load (HIV-negative participants) or CD4 and viral load testing (HIVpositive participants). Participants with positive rapid tests will have a confirmatory Western Blot assay performed and will receive HIV counseling and referrals to HIV service providers. Participants newly diagnosed with HIV at screen will be referred to community resources. Consistent with our prior trials, after obtaining the participant's permission, we will contact LINCS (Linkage, Integration, Navigation, and Comprehensive Services), a program of the San Francisco Department of Public Health (SFDPH), which provides coordinated comprehensive linkage to care, navigation and partner services for HIV-positive people living in San Francisco, particularly those who are newly HIV-positive and those who have fallen out of care.

# **Substance Use Counseling**

In addition to HIV risk-reduction counseling done at screening and month 3 visits, all participants will receive weekly 30-minute substance use counseling. This standardized protocol is based on a manualdriven psychosocial treatment program using cognitive behavioral therapy, <sup>169</sup> motivational interviewing techniques, and incorporating the Stages of Change Model. This platform has been used to treat substance use and has high acceptability among substance-using MSM. 122,173-175 Counseling will be provided by trained study staff closely supervised by a licensed clinical psychologist in weekly quality assurance session.

# **Ecological Momentary Assessments (EMA) Messages:**

As with our *Project iN* and *Better THAN* pharmacologic trials, participants will receive daily EMA texts to collect data on cocaine use patterns and medication compliance (see sample texts shown Figure 5). 163 Messages will use shorthand notations to maintain participant confidentiality. Participants will be trained on text messaging procedures and receive a reference guide during enrollment (sample guide from The Project iN Study included in the Appendix). Participants will be encouraged to regularly delete text messages and encrypt their phone with passwords for privacy. Our current studies already utilize this technology with great success and the majority of our participants prefer text appointment reminders. Moreover, text messaging has been highly acceptable in healthand research settings. 110

#### **Medical Safety and AE Assessments:**

Blood specimens will be collected via venipuncture using universal precautions. Medications taken in the 30 days prior to enrollment and while enrolled in the study will be documented. Because lorcaserin is not approved for cocaine use, we include extensive safety parameters, as is required by the Food and Drug Administration when testing a medication for a new indication. AEs and concomitant medications will be elicited from participants verbally and documented weekly. As previously noted, participants will also be given the 24-hour study phone number to communicate with the study clinician in the event of an emergency. Clinicians will follow the "Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events" (version 2.0) and UCSF IRB reporting guidelines. <sup>179</sup> Safety monitoring will include assessment, follow-up, and reporting of clinical and serious AEs, and abnormal lab results.

## **Addressing Medical/Social Needs:**

While our study will not provide direct medical care, we may identify problems and will provide referrals, identifying community providers suited for individual participants (sample list of resources referrals). Clinical staff will be available as needed for clinical consultation.


## **Qualitative Interviews:**

All participants will be scheduled for in-depth semi-structured interviews at their 12-week treatment visit. Qualitative experts, Drs. Wilson and Matheson will conduct interviews to explore participant treatment and study acceptability and assess medication adherence challenges. Semi-structured interview guides will begin with a discussion of motivations for treatment seeking and ask about the participant's history of drug use and treatment programs. The guide will then assess overall experiences as part of the study (e.g., frequency of study visits, frequency of medication dosing, appraisal of study activities and staff, study location). Participants who have experience with pharmacologic interventions for substance use treatment will be asked to compare their experiences

#### **Adverse Events**

Information regarding occurrence of adverse events will be captured throughout the study. Duration (start and stop dates and times), severity/grade, outcome, treatment and relation to study drug will be recorded on the case report form (CRF).

# 9.2 Clinical Laboratory Measurements

#### Hematology

Blood will be obtained and sent to each site's clinical hematology lab for a complete blood count (hemoglobin, hematocrit, red blood cell count, white blood cell count, white blood cell differential, and platelet count)

# **Blood Chemistry Profile**

Blood will be obtained and sent to each site's clinical chemistry lab for determination of serum sodium, potassium, chloride, bicarbonate, random glucose, BUN, creatinine, aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), alkaline phosphatase, total bilirubin, direct bilirubin, gamma-glutamyl transferase (GGT), albumin and LDH.

#### **Pregnancy Test**

A urine pregnancy test will be obtained from female subjects who are of childbearing age prior to their participation in the study.

# Urinalysis

Urine will be obtained and sent to each site's clinical laboratory for determination of cocaine metabolites (benzoylecgonine). On average, cocaine is detectable in urine for approximately 72 hours.

## 10. EVALUATIONS BY VISIT

#### 10.1 VISIT 1 (SCREENING VISIT—WEEK 1)

Review the study with the subject (subject's legal representative) and obtain written informed consent and HIPAA authorization and assent, if appropriate.

Assign the subject a unique screening number.

Record demographics data.


PI: Santos, Glenn-Milo

Record medical history, including a history of mental health, sexual behaviors and substance use, diagnosis date, and prior cocaine treatments.

Confidential

Record concomitant medications.

Perform a complete physical examination.

Collect urine sample for cocaine use and other substances test. If capable of becoming pregnant then a pregnancy test. Record results.

If urine is not positive for cocaine metabolites then place a sweat patch on participant.

# 10.2 Visit 2 (Screening Visit – week 2)

Perform and record vital signs (including weight and height for calculating BMI)

Perform and record results of blood pressure testing.

Perform and record results of ECG

Collect blood for clinical laboratory tests (chemistry, hematology, HIV test, pooled viral load test. If HIV positive, a CD4 test).

Collect and record contact information

Collect urine sample for cocaine use and other substances test. If capable of becoming pregnant then a pregnancy test. Record results.

If urine is not positive for cocaine metabolites then place a sweat patch on participant.

# **10.3** Visit 3 (Enrollment Visit – month 1)

Assign randomization. You are assigned by a computer by chance to either the lorcaserin hydrochloride or placebo groups.

Collect urine to test for cocaine metabolites and other substances.

If capable of becoming pregnant, we will collect urine and perform a pregnancy test.

Perform and record results for the BART test.

Provide study medication (lorcaserin or placebo) in medical monitoring devices ("MEMS" containers). MEMS devices will record each time you open the container to retrieve a study medication capsule.

Provided with a Wallet Card that explains that you may or may not be on a study medication (lorcaserin or placebo). This card will provide the study clinician's pager number who can provide information to other doctors in the event of an emergency. The card will also instruct the emergency room or other doctor providing treatment to provide information to the study clinician about the care they provide.

Perform ACASI questionnaire on a computer.

Meet with counselor about cocaine use.

Initiate Ecological Momentary Assessments

#### 10.4 Visit 4 (weeks 1, 2, 3, 5, 6, 7, 9, 10, and 11))

Record any Adverse Experiences and dosing compliance by downloading MEMs cap dispenser.

Meet with the counselor regarding cocaine use and use of the study medication.

Collect urine sample to test for cocaine use and other substances. If capable of becoming pregnant, we will also conduct a pregnancy test.

Answer ACASI questions on a compute


Receive the study medication: if needed, you will be given more of the study medication (except at the week 12 visit).

Meet with the study doctor or nurse: to talk about any problems with the study medication or any changes in your health or medications if needed. A physical exam may be done.

# 10.5 Visit 5 (Month 1, 2 and 3 with visit window 2 weeks before visit and 2 weeks after visit)

All the same procedures as the weekly visits **PLUS** these additional procedures:

Answer ACASI questions on a computer about your mood, your recent sexual behavior and drug use, and your feelings about being in the study.

Record any Adverse Experiences and dosing compliance.

Record changes to concomitant medications.

Perform and record results for the BART test.

Meet with the study doctor or nurse: to talk about any problems with the study medication or any changes in your health or medications if needed. A physical exam may be done.

Collect blood for clinical laboratory tests (chemistry, hematology).

At month 3 visit, collect blood for HIV test, pooled viral load test. If HIV positive, a CD4 test.

At month 3 visit, perform and record ECG results.

At month 3, perform qualitative exit interview.

#### 10.6 Early Withdrawal Visit

Record any Adverse Experiences and/or Review for adverse experiences and exclusionary medication use

Record changes to concomitant medications.

Perform complete physical examination.

Perform and record vital signs.

Collect blood for clinical laboratory tests: Chemistry, Hematology, Urinalysis, Pregnancy (urine or serum).

# 11. ADVERSE EXPERIENCE REPORTING AND DOCUMENTATION

#### 11.1 Adverse Events

An adverse event (AE) is any untoward medical occurrence in a clinical investigation of a patient administered a pharmaceutical product and that does not necessarily have a causal relationship with the treatment. An AE is therefore any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the administration of an investigational product, whether or not related to that investigational product. An unexpected AE is one of a type not identified in nature, severity, or frequency in the current Investigator's Brochure or of greater severity or frequency than expected based on the information in the Investigator's Brochure.


The Investigator will probe, via discussion with the subject, for the occurrence of AEs during each subject visit and record the information in the site's source documents. Adverse events will be recorded in the patient CRF. Adverse events will be described by duration (start and stop dates and times), severity, outcome, treatment and relation to study drug, or if unrelated, the cause.

# 11.2 AE Severity

The National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 should be used to assess and grade AE severity, including laboratory abnormalities judged to be clinically significant. The modified criteria can be found in the study manual. If the experience is not covered in the modified criteria, the guidelines shown in Table 1 below should be used to grade severity. It should be pointed out that the term "severe" is a measure of intensity and that a severe AE is not necessarily serious.

**Table 1. AE Severity Grading** 

| Severity (Toxicity Grade) | Description |
|---|---|
| Mild (1) | Transient or mild discomfort; no limitation in activity; no medical intervention or therapy required. The subject may be aware of the sign or symptom but tolerates it reasonably well. |
| Moderate (2) | Mild to moderate limitation in activity, no or minimal medical intervention/therapy required. |
| Severe (3) | Marked limitation in activity, medical intervention/therapy required, hospitalizations possible. |
| Life-threatening (4) | The subject is at risk of death due to the adverse experience as it occurred. This does not refer to an experience that hypothetically might have caused death if it were more severe. |

# **AE Relationship to Study Drug**

The relationship of an AE to the study drug should be assessed using the following the guidelines in Table 2.

Table 2. AE Relationship to Study Drug

| Relationship<br>to Drug | Comment |
|---|---|
| Definitely | Previously known toxicity of agent; or an event that follows a reasonable temporal sequence from administration of the drug; that follows a known or expected response pattern to the suspected drug; that is confirmed by stopping or reducing the dosage of the drug; and that is not explained by any other reasonable hypothesis. |
| Probably | An event that follows a reasonable temporal sequence from administration of the drug; that follows a known or expected response pattern to the suspected drug; that is confirmed by stopping or reducing the dosage of the drug; and that is unlikely to be explained by the known characteristics of the subject's clinical state or by other interventions. |


| Possibly | An event that follows a reasonable temporal sequence from administration of the drug; that follows a known or expected response pattern to that suspected drug; but that could readily have been produced by a number of other factors. |
|---|---|
| Unrelated | An event that can be determined with certainty to have no relationship to the study drug. |

# 11.3 Serious Adverse Experiences (SAE)

An SAE is defined as any AE occurring at any dose that results in any of the following outcomes:

- death
- a life-threatening adverse experience
- inpatient hospitalization or prolongation of existing hospitalization
- a persistent or significant disability/incapacity
- a congenital anomaly/birth defect

Other important medical events may also be considered an SAE when, based on appropriate medical judgment, they jeopardize the subject or require intervention to prevent one of the outcomes listed.

# 11.3 Medical Monitoring

John Walker, RN, FNP-C, research clinician, should be contacted directly at these numbers to report medical concerns or questions regarding safety.

Phone: (628) 217-6227 Pager: (415) 356-8980

Phillip Coffin, MD MIA FACP FIDSA, medical director, should be contacted directly at this number to report medical concerns or questions regarding safety.

Phone: (510) 407-2603

# 12. DISCONTINUATION AND REPLACEMENT OF SUBJECTS

# 12.1 Early Discontinuation of Study Drug

A subject may be discontinued from study treatment at any time if the subject or the investigator feels that it is not in the subject's best interest to continue. The following is a list of possible reasons for study treatment discontinuation:

- Subject withdrawal of consent (or assent)
- Subject is not compliant with study procedures
- Adverse event that in the opinion of the investigator would be in the best interest of the subject to discontinue study treatment


- Protocol violation requiring discontinuation of study treatment
- Lost to follow-up
- PI or clinician request for early termination of study
- Positive pregnancy test (females)

If a subject is withdrawn from treatment due to an adverse event, the subject will be followed and treated by the Investigator until the abnormal parameter or symptom has resolved or stabilized.

All subjects who discontinue study treatment should come in for an early discontinuation visit as soon as possible and then should be encouraged to complete all remaining scheduled visits and procedures.

All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice.

Reasonable attempts will be made by the investigator to provide a reason for subject withdrawals. The reason for the subject's withdrawal from the study will be specified in the subject's source documents Refer to Section 10 for early termination procedures.

# 12.2 Withdrawal of Subjects from the Study

A subject may be withdrawn from the study at any time if the subject or the investigator feels that it is not in the subject's best interest to continue.

All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice.

Reasonable attempts will be made by the investigator to provide a reason for subject withdrawals. The reason for the subject's withdrawal from the study will be specified in the subject's source documents. As noted above, subjects who discontinue study treatment early (i.e., they withdraw prior to Week 8 Visit ) should have an early discontinuation visit. Refer to Section 10 for early termination procedures. Subjects who withdraw after Week 8 Visit but prior to Week 12 Visit should be encouraged to come in for a final visit (and the procedures to be followed would include those for their next scheduled visit).

## 12.3 Replacement of Subjects

Subjects who withdraw from the study treatment will not be replaced.

# 13. PROTOCOL VIOLATIONS

A protocol violation occurs when the subject or investigator fails to adhere to significant protocol requirements affecting the inclusion, exclusion, subject safety and primary endpoint criteria. Protocol violations for this study include, but are not limited to, the following:

- Failure to meet inclusion/exclusion criteria
- Use of a prohibited concomitant medication (such as those listed in the exclusion criteria)

Failure to comply with Good Clinical Practice (GCP) guidelines will also result in a protocol violation. The PI will determine if a protocol violation will result in withdrawal of a subject.

When a protocol violation occurs, it will be discussed with the investigator and a Protocol Violation Form detailing the violation will be generated. This form will be signed by a Sponsor representative and the Investigator. A copy of the form will be filed in the site's regulatory binder and in the Sponsor's files.


#### 14. DATA SAFETY MONITORING

The PI along with the site physician Dr. Coffin, will be responsible for ensuring proper monitoring of the safety and efficacy of this trial, including the execution of the DSM plan, and complying with the reporting requirements, including reports to the IRB, DSMB, NIDA and (where applicable) the FDA (see Figure 1 below).



or, meets weekly to discuss all aspects of the study such as recruitment and retention, clinical or counseling issues, and any regulatory or operation issues. All study documents are monitored by the study coordinator for quality assurance on a weekly basis to ensure timely corrections to charting such as missing initials or cross-outs with error-correction. Although there is no outside monitor, the clinicians review each other's charts for accuracy, consistency, and adherence to protocol. Regular audits will be conducted as well on consent forms, laboratory logs and other data collection forms.

The interim DSMB report will contain a brief description of the trial, baseline socio-demographic characteristics of participants, retention and disposition of study participants, a description of any quality assurance or regulatory issues, a report of AEs and SAES, and the status of outcome data.

Members and affiliation: We will use the existing University of California, Los Angeles (UCLA) Data & Safety Monitoring Board for Addiction Medicine (DSMBAM), which has extensive experience in monitoring pharmacologic interventions, including among vulnerable populations. The DSMBAM has monitored all of our pharmacologic trials for substance users.

To ensure that the DSMB oversight of the study remains independent from the proposed study, the PI(Santos) as well as others who serve on the DSMBAM that might be linked with the study in some way recuse themselves from review of the present study.

The purpose of the DSMBAM is to provide oversight and monitoring of Phase I and Phase II clinical trials of pharmacological and behavioral treatments for stimulant dependence. There are three fundamental charges of the board, which are:

- To ensure the safety of trial participants
- To preserve validity and integrity of research data
- To facilitate the availability of timely as well as reliable findings to the broader clinical community

Below are members who serve as committee chairs as well as clinical research experts:


- Steven Shoptaw, PhD, is Professor in both the Department of Family Medicine and the Department of Psychiatry and Biobehavioral Sciences at UCLA. Over the past 20 years, Dr. Shoptaw has conducted a series of clinical studies in community clinic settings, primarily on topics that involve developing medical and behavioral interventions to treat substance abusers.
- Timothy M. Hall, MD, PhD, is Health Sciences Assistant Clinical Professor at UCLA Department of Family Medicine and Center for Behavioral and Addiction Medicine. His research expertise is in sexual identity formation, social/sexual MSM networks, non-gay-identified MSM, ethnography and MSM substance use.
- Gayle Baldwin, PhD, is Associate Professor in the Department of Medicine at the University of California, Los Angeles. Her research focuses on how specific immune cells fight infectious diseases and cancer.
- Dominick Frosch, PhD, is an Associate Staff Scientist in the Department of Health Services Research at the Palo Alto Medical Foundation's Research Institute. He is also an Assistant Professor of Medicine at the University of California, Los Angeles. His research is focused on developing and implementing interventions to increase patient participation in clinical decision making and understanding the effects of health information in the media on behavior.

Below are members who serve as experts in biostatistics and epidemiology:

- · Scott Comulada, PhD
- Sung-Jae Lee, PhD
- Jesse Fletcher, PhD

Below are members who serve as clinical research experts:

- · Adam Carrico, PhD
- David Farabee, PhD
- Timothy Fong, MD
- · Liz Evans, PhD
- · Lara Ray, PhD

Administrative support staff:

- Uyen Kao, MPH, Director
- Oluwadamilola O. Jolayemi, MSc, Coordinator

The DSMC evaluates known risks to subjects' participation, the safety of the subjects as pre-specified in the protocol, and monitors the operational performance of the trial. The DSMC makes recommendations to continue, amend, or terminate the trial based on their findings. Recommendations are made in writing to the study investigators. The DSMC are given blinded trial data, but may request unblinding if safety data warrant. The initial review includes a review of the following items: statement of the protocol design, characteristics of the study data collection site, inclusion/exclusion criteria, randomization plan, definition of participants (e.g., screened, enrolled, randomized, treated, drop-out, lost to follow-up), intervention definition, dosage and frequency of study drug, reasons to discontinue study or to terminate individual


participants, reasons to discontinue treatment, outcome measures, sample size target, key adherence and safety variables, and the data analysis plan.

Subsequent ongoing reviews include: enrollment data, including those screened, enrolled, and active; subject eligibility; demographic characteristics of participants (total, and by group), recruitment and retention (total and by group). Protocol compliance are evaluated by reviewing: the expected recruitment rate, study drop-outs and reasons for leaving the study, data quality assurance reports, overall data flow procedures, CRFs collected, received, and entered; protocol deviations; protocol violations; missing data; staff omissions; subject refusal to provide data; adherence to stopping rules. The data safety report are provided in total and by group, and include any relevant medical, psychosocial or laboratory data, AEs summarized in tables, individual SAE reports, concomitant medications, and concomitant illnesses. The outcome data report includes outcome data analyzed by group, masked or unblended, with or without statistical analyses, and include all outcome variables.

#### 15. STATISTICAL METHODS AND CONSIDERATIONS

Prior to the analysis of the final study data, a detailed Statistical Analysis Plan (SAP) will be written describing all analyses that will be performed. The SAP will contain any modifications to the analysis plan described below.

# 15.1 Data Sets Analyzed

All eligible patients who are randomized into the study and receive at least one dose of the study drug (the Safety Population) will be included in the safety analysis.

# 15.2 Demographic and Baseline Characteristics

The following demographic variables at screening will be summarized by treatment group: race, gender, age, educational attainment, employed, and HIV positivity.

#### 15.3 Analysis of Primary Endpoint

To establish the feasibility of enrolling and retaining 45 MSM with cocaine use disorder in a 12 week with 2:1 randomized, double-blind study of lorcaserin versus placebo. We will calculate the following feasibility measures: 1) proportion of those eligible among those screened; 2) proportion enrolled among those eligible; and 3) study completion rate. Process measures (e.g., visit length, counseling session completion) and reactions to study procedures will also be collected and reported. Betweengroup differences will be assessed using Fisher's exact and Wilcoxon rank sum tests. We will also calculate Kaplan-Meier curves for time to dropout, by group, and test for differences using the log-rank test. Precision: In the overall sample of 45, proportions will be estimated with margins of sampling error (MSEs; i.e., half widths of 95% confidence intervals) of ≤14.4 percentage points, and means with MSEs of 0.30 standard deviations, both typical for a small pilot study. While the study will only be powered to detect large between-group differences in process measures, it will provide warning of potential problems.

To explore the tolerability of lorcaserin versus placebo among MSM with cocaine use disorders, as determined by the number of adverse clinical events in the cocaine and placebo arms. We will compute the proportions of those experiencing adverse events, both overall and by type. Adverse clinical events, AEs and SAEs, and other binary safety outcomes will be presented as percent of participants that experience the safety outcome by treatment assignment. We will also classify AEs as any AE that results in stopping study medication, specific common AEs (>2% in both groups), AEs for general organ system categories, and AEs potentially related to study drug. The probability of observing at least one AE with population incidence of 1, 2, and 5% in the active arm will be 26, 45, and 70% with 2:1 randomization, respectively.


To describe the acceptability and adherence for lorcaserin versus placebo MSM with cocaine use disorders. We will measure the acceptability of lorcaserin compared to placebo among participants through a qualitative interview and survey evaluations of the study procedures, study drug characteristics, and dosing schedule at the final visit. We will determine medication adherence via MEMs Cap data, pill count, and self-report from TLFB and SMS texts. Measures of interest will include percent of doses taken, patterns of adherence, and time to stopping medication. We will assess how these measures of adherence track with patterns of cocaine use as measured in TLFB and urinalysis. Concordance of the adherence measures will be examined using weighted Kappa and correlations. Qualitative Analysis: In-depth, semi-structured qualitative interviews will be analyzed to establish the acceptability of study procedures and study medication, and identify key factors affecting treatment adherence for MSM with cocaine use disorders. Transcribed semi-structured interviews will be imported into Atlas.ti, a qualitative research software program. Data will be separated by study arm initially to determine if adherence differed between groups. If it appears there were no differences between placebo and study drug arms, then we will collapse data to assess study acceptability and adherence challenges together. If there are noticeable differences, we will analyze each set of data separately. In either scenario, we will utilize two qualitative analytic methods to interpret data. 190 First, content analysis to assess a priori themes using a structured codebook will allow us to focus on answering study questions about acceptability of study procedures and medication adherence. Second, thematic analysis primarily focused on adherence challenges will be conducted using open coding to allow themes to emerge from the data. <sup>191</sup> A coding system for the thematic analysis will be developed using an iterative process. In the initial phase, Drs. Wilson and Matheson will review transcripts and field notes to become familiar with the data, and the analytic team will make notes of their observations and potential codes for use in the initial analysis meeting. Then a thematic codebook consisting of the code definition and inclusion and exclusion criteria will be created to aid analysis. In addition to anticipated adherence challenges, additional codes will be developed independently by each analytic team member through an inductive process of identifying themes that emerge from the data. Group analysis meetings will be held to compare independently developed codes for similarity and further definition. A consensus will be reached regarding each code, its application, and definition. To ensure consistency, a codebook and dictionary will be developed with universal definitions for each code. Inter-rater reliability: The two coders will assess inter-rater reliability by calculating the correlation between a set of ratings done by two independent raters for the initial set of 3-6 transcripts, and then again on the next set of 6 transcripts. After each inter-rater reliability assessment, the codebook and codes will be revised based on reconciliation of findings done between coders. Inter-rater reliability will be assessed as a team twice during the analysis process and again at the end of analysis as a post-hoc evaluation of reliability and validity. This evolving analysis process will ensure high quality of research decisions, the rationale behind decisions, and the responsiveness of investigators to the data. 192 Once the thematic analysis codebook is developed and verified all remaining transcripts will be coded by study staff under the direction of Dr. Wilson. Further meetings will be held to discuss any differences in coding and to ensure consistency in the application of codes. Final analysis will begin with data reduction, then display, analysis and conclusion drawing using a conceptual framework in which hypothesized factors affecting adherence are assessed and unanticipated findings are identified. 193 The analytic team will work from the coded data to merge findings into a final summary and a consensus of major themes, relationships between themes, and ranking of items of most importance to adherence. This method of data reduction encompassing both site- and team-based analysis creates a robust iterative process through which the data is thoroughly discussed and analytical consensus achieved. Atlas.ti software will be used to both code and develop data displays used in the analysis

# 15.4 Analysis of Secondary Endpoints

To evaluate the *preliminary efficacy* of lorcaserin versus placebo to reduce cocaine use and HIVrelated sexual risk behaviors among MSM with cocaine use disorders, as determined by the proportion of cocaine-positivity from twice weekly urine samples and self-reported sexual behaviors. Minimum detectable effects (MDE) of the intervention on cocaine use outcomes will be substantial, as is typical of a pilot study. In our prior trial for MSM actively using stimulants, <sup>68</sup> the within-subject correlation of the repeated measures for urine positivity was 0.45, the urine positivity in the control group was 55%, and the retention was 93% at the end of the study. On this basis, we conservatively estimate that the sample will provide 80% power to detect reductions of 29 percentage points in the rate of cocaine urine positivity. In preparation for a larger trial, we will conduct exploratory assessments using GEE Poisson models to assess treatment effects on cocaine urine positivity. 194 In sensitivity analyses, we will also evaluate between-group differences on changes in: 1) any cocaine positive samples, defined as having a positive urine or sweat patch sample, over follow-up; 2) any cocaine positive samples or self-report of cocaine use in text messages; and 3) cocaine positivity from sweat samples only. Concordance of the urine testing, sweat testing, and self-reported measures will be examined using weighted Kappa and correlations. To evaluate treatment effects on cocaine-associated sexual risk behaviors, GEE Poisson, binomial, and negative binomial models will be used to assess treatment effects on HIV sexual risk behaviors including high-risk sexual behaviors while under the influence of cocaine. Findings from these analyses will be used to determine whether a linearly increasing or constant treatment effect best describes outcome patterns.

Safety and tolerability data will be summarized by treatment group.

Adverse event rates will be coded by body system and MedDra classification term. Adverse events will be tabulated by treatment group and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study drug.

# 15.5 Interim Analysis

No planned interim analysis.

#### 15.6 Sample Size and Randomization

#### 16 DATA COLLECTION, RETENTION AND MONITORING

#### 16.1 Data Collection Instruments

The Investigator will prepare and maintain adequate and accurate source documents designed to record all observations and other pertinent data for each subject treated with the study drug. Study personnel at each site will enter data from source documents corresponding to a subject's visit into the protocol-specific paper CRF when the information corresponding to that visit is available. Staff will upload data to the eCRF. Subjects will not be identified by name in the study database or on any study documents to be collected, but will be identified by subject number and date.


For eCRFs: If a correction is required for an eCRF, the time and date stamps track the person entering or updating eCRF data and creates an electronic audit trail. For paper CRFs: If a correction is made on a CRF, the study staff member will line through the incorrect data, write in the correct data and initial and date the change.

The Investigator is responsible for all information collected on subjects enrolled in this study. All data collected during the course of this study must be reviewed and verified for completeness and accuracy by the Investigator. A copy of the CRF will remain at the Investigator's site at the completion of the study.

# **16.2 Data Management Procedures**

The data will be entered into a validated database. The Data Management group will be responsible for data processing, in accordance with procedural documentation. Database lock will occur once quality assurance procedures have been completed.

All procedures for the handling and analysis of data will be conducted using good computing practices meeting FDA guidelines for the handling and analysis of data for clinical trials.

# 16.3 Data Quality Control and Reporting

After data have been entered into the study database, a system of computerized data validation checks will be implemented and applied to the database on a regular basis. *For paper studies:* Query reports (Data Clarification Requests) pertaining to data omissions and discrepancies will be forwarded to the Investigators and study monitors for resolution. The study database will be updated in accordance with the resolved queries. All changes to the study database will be documented.

## 16.4 Archival of Data

The database is safeguarded against unauthorized access by established security procedures; appropriate backup copies of the database and related software files will be maintained. Databases are backed up by the database administrator in conjunction with any updates or changes to the database.

At critical junctures of the protocol (e.g., production of interim reports and final reports), data for analysis is locked and cleaned per established procedures.

# 16.5 Availability and Retention of Investigational Records

The Investigator must make study data accessible to the monitor, other authorized representatives of the Sponsor (or designee), IRB, and Regulatory Agency (e.g., FDA) inspectors upon request. A file for each subject must be maintained that includes the signed Informed Consent, HIPAA Authorization and Assent Form and copies of all source documentation related to that subject. The Investigator must ensure the reliability and availability of source documents from which the information on the CRF was derived.

All study documents (patient files, signed informed consent forms, copies of CRFs, Study File Notebook, etc.) must be kept secured for a period of two years following marketing of the investigational product or for two years after centers have been notified that the IND has been discontinued. There may be other circumstances for which the Sponsor is required to maintain


study records and, therefore, the Sponsor should be contacted prior to removing study records for any reason.

## 16.6 Monitoring

Monitoring visits will be conducted by representatives of the Sponsor according to the U.S. CFR Title 21 Parts 50, 56, and 312 and ICH Guidelines for GCP (E6). By signing this protocol, the Investigator grants permission to the Sponsor (or designee), and appropriate regulatory authorities to conduct on-site monitoring and/or auditing of all appropriate study documentation.

# 16.7 Subject Confidentiality

In order to maintain subject confidentiality, only a subject number and subject initials will identify all study subjects on CRFs and other documentation submitted to the Sponsor. Additional subject confidentiality issues (if applicable) are covered in the Clinical Study Agreement.

# 17 ADMINISTRATIVE, ETHICAL, REGULATORY CONSIDERATIONS

The study will be conducted according to the Declaration of Helsinki, Protection of Human Volunteers (21 CFR 50), Institutional Review Boards (21 CFR 56), and Obligations of Clinical Investigators (21 CFR 312).

To maintain confidentiality, all laboratory specimens, evaluation forms, reports and other records will be identified by a coded number and initials only. All study records will be kept in a locked file cabinet and code sheets linking a patient's name to a patient identification number will be stored separately in another locked file cabinet. Clinical information will not be released without written permission of the subject, except as necessary for monitoring by the FDA. The Investigator must also comply with all applicable privacy regulations (e.g., Health Insurance Portability and Accountability Act of 1996, EU Data Protection Directive 95/46/EC).

#### 17.1 Protocol Amendments

Any amendment to the protocol will be written by the Principal Investigator. Protocol amendments cannot be implemented without prior written IRB approval except as necessary to eliminate immediate safety hazards to patients. A protocol amendment intended to eliminate an apparent immediate hazard to patients may be implemented immediately, provided the IRBs are notified within five working days.

#### 17.2 Institutional Review Boards

The protocol and consent form will be reviewed and approved by the IRB of each participating center prior to study initiation. Serious adverse experiences regardless of causality will be reported to the IRB/IEC in accordance with the standard operating procedures and policies of the IRB/IEC, and the Investigator will keep the IRB/IEC informed as to the progress of the study. The Investigator will obtain assurance of IRB/IEC compliance with regulations.

Any documents that the IRB/IEC may need to fulfill its responsibilities (such as protocol, protocol amendments, Investigator's Brochure, consent forms, information concerning patient recruitment, payment or compensation procedures, or other pertinent information) will be submitted to the IRB/IEC. The IRB/IECs written unconditional approval of the study protocol


and the informed consent form will be in the possession of the Investigator before the study is initiated. The IRB/IECs unconditional approval statement will be transmitted by the Investigator to prior to the shipment of study supplies to the site. This approval must refer to the study by exact protocol title and number and should identify the documents reviewed and the date of review.

Protocol and/or informed consent modifications or changes may not be initiated without prior written IRB approval except when necessary to eliminate immediate hazards to the patients or when the change(s) involves only logistical or administrative aspects of the study. Such modifications will be submitted to the IRB and written verification that the modification was submitted and subsequently approved should be obtained.

The IRB must be informed of revisions to other documents originally submitted for review; serious and/or unexpected adverse experiences occurring during the study in accordance with the standard operating procedures and policies of the IRB; new information that may affect adversely the safety of the patients of the conduct of the study; an annual update and/or request for re-approval; and when the study has been completed.

#### 17.3 Informed Consent Form

Informed consent will be obtained in accordance with the Declaration of Helsinki, ICH GCP, US Code of Federal Regulations for Protection of Human Subjects (21 CFR 50.25[a,b], CFR 50.27, and CFR Part 56, Subpart A), the Health Insurance Portability and Accountability Act (HIPAA, if applicable), and local regulations.

The Investigator will prepare the informed consent form, assent and HIPAA authorization and provide the documents to the Sponsor or designee for approval prior to submission to the IRB/IEC. The consent form generated by the Investigator must be acceptable to the Sponsor and be approved by the IRB. The written consent document will embody the elements of informed consent as described in the International Conference on Harmonisation and will also comply with local regulations. The Investigator will send an IRB-approved copy of the Informed Consent Form to the Sponsor (or designee) for the study file.

A properly executed, written, informed consent will be obtained from each subject prior to entering the subject into the trial. Information should be given in both oral and written form and subjects (or their legal representatives) must be given ample opportunity to inquire about details of the study. If appropriate and required by the local IRB, assent from the subject will also be obtained. If a subject is unable to sign the informed consent form (ICF) and the HIPAA authorization, a legal representative may sign for the subject. A copy of the signed consent form (and assent) will be given to the subject or legal representative of the subject and the original will be maintained with the subject's records.

#### 17.4 Publications

The preparation and submittal for publication of manuscripts containing the study results shall be in accordance with a process determined by mutual written agreement among the Principal Investigator and participating institutions. The publication or presentation of any study results shall comply with all applicable privacy laws, including, but not limited to, the Health Insurance Portability and Accountability Act of 1996.

#### 17.5 Investigator Responsibilities

By signing the Agreement of Investigator form, the Investigator agrees to:

1. Conduct the study in accordance with the protocol and only make changes after notifying the Sponsor (or designee), except when to protect the safety, rights or welfare of subjects.


- 2. Personally conduct or supervise the study (or investigation).
- 3. Ensure that the requirements relating to obtaining informed consent and IRB review and approval meet federal guidelines, as stated in § 21 CFR, parts 50 and 56.
- 4. Report to the Sponsor or designee any AEs that occur in the course of the study, in accordance with §21 CFR 312.64.
- 5. Ensure that all associates, colleagues and employees assisting in the conduct of the study are informed about their obligations in meeting the above commitments.
- 6. Maintain adequate and accurate records in accordance with §21 CFR 312.62 and to make those records available for inspection with the Sponsor (or designee).
- 7. Ensure that an IRB that complies with the requirements of §21 CFR part 56 will be responsible for initial and continuing review and approval of the clinical study.
- 8. Promptly report to the IRB and the Sponsor (or designee) all changes in the research activity and all unanticipated problems involving risks to subjects or others (to include amendments and IND safety reports).
- 9. Seek IRB approval before any changes are made in the research study, except when necessary to eliminate hazards to the patients/subjects.
- 10. Comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements listed in § 21 CFR part 312.


#### 18 APPENDICES

# **Appendix 1: Study Procedures**

| Table 2. The TLC Study<br>Procedures | Enr | Wk | Bi-<br>wk | Dly | M 1&2 | M 3 |
|---|---|---|---|---|---|---|
| Informed consent | | | | | | |
| Safety lab assessment | | | | | X | X |
| Rapid HIV test*, CD4, viral load | | | | | | X |
| HIV risk reduction counseling | | | | | | X |
| Medical history and SCID | | | | | | |
| Vital signs, weight | X | | | | X | X |
| Physical exam | X | | | | | X |
| Medication Training | X | | | | | |
| Randomization | X | | | | | |
| Urine testing for cocaine | X | X | X | | X | X |
| Sweat patch testing for cocaine | X | X | | | X | X |
| CAPI assessments | X | X | | | X | X |
| AE assessments | | X | | | X | X |
| Substance use counseling | | X | | | | |
| Qualitative Interviews | | | | | | X |
| Text Messaging | | | | X | | |
| Notes: *Confirmatory HIV testing will be performed for reactive tests. Scr=Screening, Enr=Enrollment, Wk=Weekly, Bi-wk=Biweekly/twice weekly, Dly=Daily, M=Monthly | | | | | | |

# 18.2 Appendix 2: References:

- 1. Riezzo I, Fiore C, De Carlo D, et al. Side effects of cocaine abuse: multiorgan toxicity and pathological consequences. Curr Med Chem 2012;19:5624-46.
- 2. Karila L, Petit A, Lowenstein W, Reynaud M. Diagnosis and consequences of cocaine addiction. Curr Med Chem 2012;19:5612-8.
- 3. Substance Abuse and Mental Health Services Administration. Drug Abuse Warning Network, 2011: National Estimates of Drug-Related Emergency Department Visits Rockville, MD: HHS; 2013 04/14/2014.
- 4. United Nations Office on Drugs and Crime. World Drug Report 2009. Vienna, Austria 2009.
- 5. Degenhardt L, Chiu WT, Sampson N, et al. Toward a global view of alcohol, tobacco, cannabis, and cocaine use: findings from the WHO World Mental Health Surveys. PLoS Med 2008;5:e141.
- 6. Anthony J, Warner L, Kessler R. Comparative epidemiology of dependence on tobacco, alcohol, controlled substances, and inhalants: Basic findings from the National Comorbidity Survey. Experimental and Clinical Psychopharmacology 1994;23:244.
- 7. Degenhardt L, Baxter AJ, Lee YY, et al. The global epidemiology and burden of psychostimulant dependence: Findings from the Global Burden of Disease Study 2010. Drug Alcohol Depend 2014.
- 8. Drugs of Abuse Sweat Patch. 2013. (Accessed 12/20/14, 2014, at http://www.pharmchem.com/default.asp?page=2.25.)
- 9. Vandhuick O, Pistorius MA, Jousse S, et al. [Drug addiction and cardiovascular pathologies]. Journal des maladies vasculaires 2004;29:243-8.
- 10. Kloner RA, Hale S, Alker K, Rezkalla S. The effects of acute and chronic cocaine use on the heart. Circulation 1992;85:407-19.

Version 2 Version Date: 7/22/2017 

- 11. McCord J, Jneid H, Hollander JE, et al. Management of cocaine-associated chest pain and myocardial infarction: a scientific statement from the American Heart Association Acute Cardiac Care Committee of the Council on Clinical Cardiology. Circulation 2008;117:1897-907.
- 12. Phillips K, Luk A, Soor GS, Abraham JR, Leong S, Butany J. Cocaine cardiotoxicity: a review of the pathophysiology, pathology, and treatment options. American journal of cardiovascular drugs: drugs, devices, and other interventions 2009;9:177-96.
- 13. Steinhauer JR, Caulfield JB. Spontaneous coronary artery dissection associated with cocaine use: a case report and brief review. Cardiovascular pathology: the official journal of the Society for Cardiovascular Pathology 2001;10:141-5.
- 14. Sanchez T, Finlayson T, Drake A, et al. Human immunodeficiency virus (HIV) risk, prevention, and testing behaviors--United States, National HIV Behavioral Surveillance System: men who have sex with men, November 2003-April 2005. MMWR Surveill Summ 2006;55:1-16.
- 15. SAMHSA. National Survey on Drug Use and Health. Office of Applied Studies 2004.
- 16. Raymond HF. Estimated number of stimulant using men-who-have-sex-with-men in San Francisco. In: Santos GM, ed. San Francisco, CA2012.
- 17. Raymond HF. National HIV Behavioral Surveillance MSM cycle 4 stimulant use data In: Santos GM, ed. San Francisco, CA2014.
- 18. Raymond HF, Chen YH, Ick T, et al. A new trend in the HIV epidemic among men who have sex with men, San Francisco, 2004-2011. J Acquir Immune Defic Syndr 2013;62:584-9.
- 19. San Francisco Department of Public Health. 2012 HIV/AIDS Epidemiology Annual Report. San Francisco San Francisco Department of Public Health 2013.
- 20. San Francisco Department of Public Health. 2013 HIV/AIDS Epidemiology Annual Report. San Francisco San Francisco Department of Public Health 2014.
- 21. Prejean J, Song R, Hernandez A, et al. Estimated HIV incidence in the United States, 2006-2009. PLoS One 2011;6:e17502.
- 22. Hall HI, Song R, Rhodes P, et al. Estimation of HIV incidence in the United States. Jama 2008;300:520-9.
- 23. Purcell D, Johnson C, Lansky A, et al. Calculating HIV and Syphilis Rates for Risk Groups: Estimating the National Population Size of Men Who Have Sex with Men. National STD Prevention Conference. Atlanta, GA 2010.
- 24. San Francisco Department of Public Health. 2010 HIV/AIDS Epidemiology Annual Report. San Francisco San Francisco Department of Public Health 2011.
- 25. ONAP. National HIV/AIDS Strategy for the United States. In: Policy TWHOoNA, ed. Washington, DC2010.
- 26. Volkow ND, Wang GJ, Fowler JS, Telang F, Jayne M, Wong C. Stimulant-induced enhanced sexual desire as a potential contributing factor in HIV transmission. Am J Psychiatry 2007:164:157-60.
- 27. Colfax G, Coates TJ, Husnik MJ, et al. Longitudinal patterns of methamphetamine, popper (amyl nitrite), and cocaine use and high-risk sexual behavior among a cohort of san francisco men who have sex with men. J Urban Health 2005;82:i62-70.
- 28. Shoptaw S, Reback CJ, Frosch DL, Rawson RA. Stimulant abuse treatment as HIV prevention. J Addict Dis 1998;17:19-32.
- 29. Celentano DD, Valleroy LA, Sifakis F, et al. Associations between substance use and sexual risk among very young men who have sex with men. Sex Transm Dis 2006;33:265-71.
- 30. Melis MR, Argiolas A. Dopamine and sexual behavior. Neurosci Biobehav Rev 1995;19:19-38.
- 31. Cunningham KA, Anastasio NC. Serotonin at the nexus of impulsivity and cue reactivity in cocaine addiction. Neuropharmacology 2014;76 Pt B:460-78.
- 32. Winhusen T, Lewis D, Adinoff B, et al. Impulsivity is associated with treatment non-completion in cocaine- and methamphetamine-dependent patients but differs in nature as a function of stimulant-dependence diagnosis. J Subst Abuse Treat 2013;44:541-7.


- 33. McKirnan DJ, Ostrow DG, Hope B. Sex, drugs and escape: a psychological model of HIV-risk sexual behaviours. AIDS Care 1996;8:655-69.
- 34. Lejuez CW, Bornovalova MA, Daughters SB, Curtin JJ. Differences in impulsivity and sexual risk behavior among inner-city crack/cocaine users and heroin users. Drug Alcohol Depend 2005;77:169-75.
- 35. Parsons JT, Halkitis PN. Sexual and drug-using practices of HIV-positive men who frequent public and commercial sex environments. AIDS Care 2002;14:815-26.
- 36. Purcell DW, Parsons JT, Halkitis PN, Mizuno Y, Woods WJ. Substance use and sexual transmission risk behavior of HIV-positive men who have sex with men. J Subst Abuse 2001;13:185-200.
- 37. Mansergh G, Colfax GN, Marks G, Rader M, Guzman R, Buchbinder S. The Circuit Party Men's Health Survey: findings and implications for gay and bisexual men. Am J Public Health 2001;91:953-8.
- 38. Mimiaga MJ, Reisner SL, Fontaine YM, et al. Walking the line: stimulant use during sex and HIV risk behavior among Black urban MSM. Drug Alcohol Depend 2010;110:30-7.
- 39. Colfax G, Vittinghoff E, Husnik MJ, et al. Substance use and sexual risk: a participant- and episode-level analysis among a cohort of men who have sex with men. Am J Epidemiol 2004;159:1002-12.
- 40. Ober A, Shoptaw S, Wang PC, Gorbach P, Weiss RE. Factors associated with event-level stimulant use during sex in a sample of older, low-income men who have sex with men in Los Angeles. Drug Alcohol Depend 2009;102:123-9.
- 41. Mackesy-Amiti ME, Fendrich M, Johnson TP. Symptoms of substance dependence and risky sexual behavior in a probability sample of HIV-negative men who have sex with men in Chicago. Drug Alcohol Depend 2010;110:38-43.
- 42. Lambert G, Cox J, Hottes TS, et al. Correlates of unprotected anal sex at last sexual episode: analysis from a surveillance study of men who have sex with men in Montreal. AIDS Behav 2011;15:584-95.
- 43. Bowers JR, Branson CM, Fletcher JB, Reback CJ. Predictors of HIV Sexual Risk Behavior among Men Who Have Sex with Men, Men Who Have Sex with Men and Women, and Transgender Women. Int J Sex Health 2012;24:290-302.
- 44. Santos GM, Coffin PO, Das M, et al. Dose-response associations between number and frequency of substance use and high-risk sexual behaviors among HIV-negative substance-using men who have sex with men (SUMSM) in San Francisco. J Acquir Immune Defic Syndr 2013;63:540-4.
- 45. Ostrow DG, Plankey MW, Cox C, et al. Specific sex drug combinations contribute to the majority of recent HIV seroconversions among MSM in the MACS. J Acquir Immune Defic Syndr 2009;51:349-55.
- 46. Koblin BA, Husnik MJ, Colfax G, et al. Risk factors for HIV infection among men who have sex with men. AIDS 2006;20:731-9.
- 47. Ostrow DG, DiFranceisco WJ, Chmiel JS, Wagstaff DA, Wesch J. A case-control study of human immunodeficiency virus type 1 seroconversion and risk-related behaviors in the Chicago MACS/CCS Cohort, 1984-1992. Multicenter AIDS Cohort Study. Coping and Change Study. Am J Epidemiol 1995;142:875-83.
- 48. Carrico AW, Pollack LM, Stall RD, et al. Psychological processes and stimulant use among men who have sex with men. Drug Alcohol Depend 2012;123:79-83.
- 49. Hinkin CH, Barclay TR, Castellon SA, et al. Drug use and medication adherence among HIV-1 infected individuals. AIDS Behav 2007;11:185-94.
- 50. Carrico AW. Substance use and HIV disease progression in the HAART era: implications for the primary prevention of HIV. Life Sci 2011;88:940-7.


- 51. Shoptaw S, Stall R, Bordon J, et al. Cumulative exposure to stimulants and immune function outcomes among HIV-positive and HIV-negative men in the Multicenter AIDS Cohort Study. Int J STD AIDS 2012;23:576-80.
- 52. Cook JA, Burke-Miller JK, Cohen MH, et al. Crack cocaine, disease progression, and mortality in a multicenter cohort of HIV-1 positive women. AIDS 2008;22:1355-63.
- 53. Carrico AW, Johnson MO, Morin SF, et al. Stimulant use is associated with immune activation and depleted tryptophan among HIV-positive persons on anti-retroviral therapy. Brain Behav Immun 2008;22:1257-62.
- 54. Roth MD, Tashkin DP, Choi R, Jamieson BD, Zack JA, Baldwin GC. Cocaine enhances human immunodeficiency virus replication in a model of severe combined immunodeficient mice implanted with human peripheral blood leukocytes. J Infect Dis 2002;185:701-5.
- 55. Bagasra O, Pomerantz RJ. Human immunodeficiency virus type 1 replication in peripheral blood mononuclear cells in the presence of cocaine. J Infect Dis 1993;168:1157-64.
- 56. Cohen MS, Chen YQ, McCauley M, et al. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med 2011;365:493-505.
- 57. Santos GM, Das M, Colfax GN. Interventions for non-injection substance use among US men who have sex with men: what is needed. AIDS Behav 2011;15 Suppl 1:S51-6.
- 58. Mackesy-Amiti ME, Fendrich M, Johnson TP. Substance-related problems and treatment among men who have sex with men in comparison to other men in Chicago. J Subst Abuse Treat 2009;36:227-33.
- 59. Shallow S. Persons attending substance abuse treatment programs. San Francisco, CA: San Francisco Department of Public Health; 2004.
- 60. Santos GM, Coffin PO, Vittinghoff E, et al. Substance use and drinking outcomes in Personalized Cognitive Counseling randomized trial for episodic substance-using men who have sex with men. Drug Alcohol Depend 2014;138:234-9.
- 61. Coffin PO, Santos GM, Colfax G, et al. Adapted Personalized Cognitive Counseling for Episodic Substance-Using Men Who Have Sex with Men: A Randomized Controlled Trial. AIDS Behav 2014.
- 62. Dutra L, Stathopoulou G, Basden SL, Leyro TM, Powers MB, Otto MW. A meta-analytic review of psychosocial interventions for substance use disorders. Am J Psychiatry 2008;165:179-87.
- 63. Kampman KM. The search for medications to treat stimulant dependence. Addict Sci Clin Pract 2008;4:28-35.
- 64. Alvarez Y, Perez-Mana C, Torrens M, Farre M. Antipsychotic drugs in cocaine dependence: a systematic review and meta-analysis. J Subst Abuse Treat 2013;45:1-10.
- 65. Jorenby DE, Leischow SJ, Nides MA, et al. A controlled trial of sustained-release bupropion, a nicotine patch, or both for smoking cessation. N Engl J Med 1999;340:685-91.
- 66. Fiellin DA. Substance use and disorders in HIV-infected patients: Impact and new treatment strategies. Top HIV Med 2004;12:77-82.
- 67. Johnson RE, Chutuape MA, Strain EC, Walsh SL, Stitzer ML, Bigelow GE. A comparison of levomethadyl acetate, buprenorphine, and methadone for opioid dependence. N Engl J Med 2000;343:1290-7.
- 68. Colfax GN, Santos GM, Das M, et al. Mirtazapine to reduce methamphetamine use: a randomized controlled trial. Arch Gen Psychiatry 2011;68:1168-75.
- 69. Rothman RB, Blough BE, Baumann MH. Dopamine/serotonin releasers as medications for stimulant addictions. Prog Brain Res 2008;172:385-406.
- 70. Higgins GA, Sellers EM, Fletcher PJ. From obesity to substance abuse: therapeutic opportunities for 5-HT2C receptor agonists. Trends Pharmacol Sci 2013;34:560-70.
- 71. Alex KD, Pehek EA. Pharmacologic mechanisms of serotonergic regulation of dopamine neurotransmission. Pharmacol Ther 2007;113:296-320.


- 72. Di Matteo V, Di Giovanni G, Di Mascio M, Esposito E. SB 242084, a selective serotonin2C receptor antagonist, increases dopaminergic transmission in the mesolimbic system. Neuropharmacology 1999;38:1195-205.
- 73. Anastasio NC, Liu S, Maili L, et al. Variation within the serotonin (5-HT) 5-HT2C receptor system aligns with vulnerability to cocaine cue reactivity. Transl Psychiatry 2014;4:e369.
- 74. Anastasio NC, Stutz SJ, Fox RG, et al. Functional status of the serotonin 5-HT2C receptor (5-HT2CR) drives interlocked phenotypes that precipitate relapse-like behaviors in cocaine dependence. Neuropsychopharmacology 2014;39:370-82.
- 75. Bubar MJ, Cunningham KA. Serotonin 5-HT2A and 5-HT2C receptors as potential targets for modulation of psychostimulant use and dependence. Curr Top Med Chem 2006;6:1971-85.
- 76. Bubar MJ, Cunningham KA. Prospects for serotonin 5-HT2R pharmacotherapy in psychostimulant abuse. Prog Brain Res 2008;172:319-46.
- 77. Burton CL, Rizos Z, Diwan M, Nobrega JN, Fletcher PJ. Antagonizing 5-HT(2)A receptors with M100907 and stimulating 5-HT(2)C receptors with Ro60-0175 blocks cocaine-induced locomotion and zif268 mRNA expression in Sprague-Dawley rats. Behavioural brain research 2013:240:171-81.
- 78. Craige CP, Unterwald EM. Serotonin (2C) receptor regulation of cocaine-induced conditioned place preference and locomotor sensitization. Behavioural brain research 2013;238:206-10.
- 79. Cunningham KA, Fox RG, Anastasio NC, et al. Selective serotonin 5-HT(2C) receptor activation suppresses the reinforcing efficacy of cocaine and sucrose but differentially affects the incentive-salience value of cocaine- vs. sucrose-associated cues. Neuropharmacology 2011;61:513-23.
- 80. Filip M, Alenina N, Bader M, Przegalinski E. Behavioral evidence for the significance of serotoninergic (5-HT) receptors in cocaine addiction. Addict Biol 2010;15:227-49.
- 81. Filip M, Spampinato U, McCreary AC, Przegalinski E. Pharmacological and genetic interventions in serotonin (5-HT)(2C) receptors to alter drug abuse and dependence processes. Brain Res 2012;1476:132-53.
- 82. Katsidoni V, Apazoglou K, Panagis G. Role of serotonin 5-HT2A and 5-HT2C receptors on brain stimulation reward and the reward-facilitating effect of cocaine. Psychopharmacology (Berl) 2011;213:337-54.
- 83. Leggio GM, Cathala A, Moison D, Cunningham KA, Piazza PV, Spampinato U. Serotonin2C receptors in the medial prefrontal cortex facilitate cocaine-induced dopamine release in the rat nucleus accumbens. Neuropharmacology 2009;56:507-13.
- 84. Manvich DF, Kimmel HL, Howell LL. Effects of serotonin 2C receptor agonists on the behavioral and neurochemical effects of cocaine in squirrel monkeys. J Pharmacol Exp Ther 2012;341:424-34.
- 85. Pockros LA, Pentkowski NS, Conway SM, Ullman TE, Zwick KR, Neisewander JL. 5-HT(2A) receptor blockade and 5-HT(2C) receptor activation interact to reduce cocaine hyperlocomotion and Fos protein expression in the caudate-putamen. Synapse 2012;66:989-1001.
- 86. Thomsen WJ, Grottick AJ, Menzaghi F, et al. Lorcaserin, a novel selective human 5-hydroxytryptamine2C agonist: in vitro and in vivo pharmacological characterization. J Pharmacol Exp Ther 2008;325:577-87.
- 87. Grottick AJ, Fletcher PJ, Higgins GA. Studies to investigate the role of 5-HT(2C) receptors on cocaine- and food-maintained behavior. J Pharmacol Exp Ther 2000;295:1183-91.
- 88. Pelloux Y, Dilleen R, Economidou D, Theobald D, Everitt BJ. Reduced forebrain serotonin transmission is causally involved in the development of compulsive cocaine seeking in rats. Neuropsychopharmacology 2012;37:2505-14.
- 89. Kohut S, Bergman J, Mello N. Pretreatment with either a 5-HT2C agonist or 5-HT2A antagonist decreases cocaine self-administration. The FASEB Journal 2014;28.


- 90. Cunningham KA, Anastasio NC, Fox RG, et al. Synergism between a serotonin 5-HT2A receptor (5-HT2AR) antagonist and 5-HT2CR agonist suggests new pharmacotherapeutics for cocaine addiction. ACS Chem Neurosci 2013;4:110-21.
- 91. Neisewander JL, Acosta JI. Stimulation of 5-HT2C receptors attenuates cue and cocaine-primed reinstatement of cocaine-seeking behavior in rats. Behav Pharmacol 2007;18:791-800.
- 92. Fletcher PJ, Tampakeras M, Sinyard J, Slassi A, Isaac M, Higgins GA. Characterizing the effects of 5-HT(2C) receptor ligands on motor activity and feeding behaviour in 5-HT(2C) receptor knockout mice. Neuropharmacology 2009;57:259-67.
- 93. Fletcher PJ, Rizos Z, Sinyard J, Tampakeras M, Higgins GA. The 5-HT2C receptor agonist Ro60-0175 reduces cocaine self-administration and reinstatement induced by the stressor yohimbine, and contextual cues. Neuropsychopharmacology 2008;33:1402-12.
- 94. Burbassi S, Cervo L. Stimulation of serotonin2C receptors influences cocaine-seeking behavior in response to drug-associated stimuli in rats. Psychopharmacology (Berl) 2008;196:15-27.
- 95. Levin ED, Johnson JE, Slade S, et al. Lorcaserin, a 5-HT2C agonist, decreases nicotine self-administration in female rats. J Pharmacol Exp Ther 2011;338:890-6.
- 96. Higgins GA, Silenieks LB, Rossmann A, et al. The 5-HT2C receptor agonist lorcaserin reduces nicotine self-administration, discrimination, and reinstatement: relationship to feeding behavior and impulse control. Neuropsychopharmacology 2012;37:1177-91.
- 97. Volkow ND, Wise RA. How can drug addiction help us understand obesity? Nat Neurosci 2005;8:555-60.
- 98. Kenny PJ. Common cellular and molecular mechanisms in obesity and drug addiction. Nat Rev Neurosci 2011;12:638-51.
- 99. Volkow ND, O'Brien CP. Issues for DSM-V: should obesity be included as a brain disorder? Am J Psychiatry 2007;164:708-10.
- 100. Higgins GA, Silenieks LB, Lau W, et al. Evaluation of chemically diverse 5-HT(2)c receptor agonists on behaviours motivated by food and nicotine and on side effect profiles. Psychopharmacology (Berl) 2013;226:475-90.
- 101. Fletcher PJ, Rizos Z, Noble K, Higgins GA. Impulsive action induced by amphetamine, cocaine and MK801 is reduced by 5-HT(2C) receptor stimulation and 5-HT(2A) receptor blockade. Neuropharmacology 2011;61:468-77.
- 102. Navarra R, Comery TA, Graf R, Rosenzweig-Lipson S, Day M. The 5-HT(2C) receptor agonist WAY-163909 decreases impulsivity in the 5-choice serial reaction time test. Behavioural brain research 2008;188:412-5.
- 103. Chan EW, He Y, Chui CS, Wong AY, Lau WC, Wong IC. Efficacy and safety of lorcaserin in obese adults: a meta-analysis of 1-year randomized controlled trials (RCTs) and narrative review on short-term RCTs. Obes Rev 2013;14:383-92.
- 104. Belviq (lorcaserin HCl) Prescribing Information 2012. (Accessed April 16, 2014, 2014, at http://www.belviq.com/documents/Belviq Prescribing information.pdf.)
- 105. Smith SR, Weissman NJ, Anderson CM, et al. Multicenter, placebo-controlled trial of lorcaserin for weight management. N Engl J Med 2010;363:245-56.
- 106. Fidler MC, Sanchez M, Raether B, et al. A one-year randomized trial of lorcaserin for weight loss in obese and overweight adults: the BLOSSOM trial. J Clin Endocrinol Metab 2011;96:3067-77.
- 107. O'Neil PM, Smith SR, Weissman NJ, et al. Randomized placebo-controlled clinical trial of lorcaserin for weight loss in type 2 diabetes mellitus: the BLOOM-DM study. Obesity (Silver Spring) 2012;20:1426-36.
- 108. Shram MJ, Schoedel KA, Bartlett C, Shazer RL, Anderson CM, Sellers EM. Evaluation of the abuse potential of lorcaserin, a serotonin 2C (5-HT2C) receptor agonist, in recreational polydrug users. Clin Pharmacol Ther 2011;89:683-92.


- 109. Jenkins RA. Recruiting substance-using men who have sex with men into HIV prevention research: current status and future directions. AIDS Behav 2012;16:1411-9.
- 110. Armstrong AW, Watson AJ, Makredes M, Frangos JE, Kimball AB, Kvedar JC. Text-message reminders to improve sunscreen use: a randomized, controlled trial using electronic monitoring. Arch Dermatol 2009;145:1230-6.
- 111. Cocosila M, Archer N, Haynes RB, Yuan Y. Can wireless text messaging improve adherence to preventive activities? Results of a randomised controlled trial. Int J Med Inform 2009;78:230-8.
- 112. Franklin VL, Waller A, Pagliari C, Greene SA. A randomized controlled trial of Sweet Talk, a text-messaging system to support young people with diabetes. Diabet Med 2006;23:1332-8.
- 113. Granholm E, Ben-Zeev D, Link PC, Bradshaw KR, Holden JL. Mobile Assessment and Treatment for Schizophrenia (MATS): A Pilot Trial of An Interactive Text-Messaging Intervention for Medication Adherence, Socialization, and Auditory Hallucinations. Schizophr Bull 2011.
- 114. Miloh T, Annunziato R, Arnon R, et al. Improved adherence and outcomes for pediatric liver transplant recipients by using text messaging. Pediatrics 2009;124:e844-50.
- 115. Petrie KJ, Perry K, Broadbent E, Weinman J. A text message programme designed to modify patients' illness and treatment beliefs improves self-reported adherence to asthma preventer medication. Br J Health Psychol 2011.
- 116. Rodgers A, Corbett T, Bramley D, et al. Do u smoke after txt? Results of a randomised trial of smoking cessation using mobile phone text messaging. Tob Control 2005;14:255-61.
- 117. Shapiro JR, Bauer S, Andrews E, et al. Mobile therapy: Use of text-messaging in the treatment of bulimia nervosa. Int J Eat Disord 2010;43:513-9.
- 118. Wei J, Hollin I, Kachnowski S. A review of the use of mobile phone text messaging in clinical and healthy behaviour interventions. J Telemed Telecare 2011;17:41-8.
- 119. McClure JB, Swan GE, St John J, et al. Pharmacogenetic smoking cessation intervention in a health care setting: a pilot feasibility study. Nicotine & tobacco research: official journal of the Society for Research on Nicotine and Tobacco 2013;15:518-26.
- 120. Gonseth S, Abarca M, Madrid C, Cornuz J. A pilot study combining individual-based smoking cessation counseling, pharmacotherapy, and dental hygiene intervention. BMC public health 2010;10:348.
- 121. Stall R, Purcell D. Intertwining epidemics: A review of research on substance use among men who have sex with men and its connection to the AIDS epidemic. AIDS and Behavior 2000;4:181-92.
- 122. Das M, Santos D, Matheson T, et al. Feasibility and acceptability of a phase II randomized pharmacologic intervention for methamphetamine dependence in high-risk men who have sex with men. AIDS 2010;24:991-1000.
- 123. Coffin PO, Santos GM, Das M, et al. Aripiprazole for the treatment of methamphetamine dependence: a randomized, double-blind, placebo-controlled trial. Addiction 2013;108:751-61.
- 124. Das M, Dadasovich R, Matheson T, et al. Adapting an Effective HIV Prevention Intervention, Personalized Cognitive Counseling, for Episodic Substance-Using Men who have Sex with Men (SUMSM). XVIII International AIDS Conference. Vienna, Austria. Abstract #WEPE03242010.
- 125. Mansergh G, Koblin BA, McKirnan DJ, et al. An intervention to reduce HIV risk behavior of substance-using men who have sex with men: a two-group randomized trial with a nonrandomized third group. PLoS Med 2010;7:e1000329.
- 126. Fuqua V, Chen YH, Packer T, et al. Using social networks to reach Black MSM for HIV testing and linkage to care. AIDS Behav 2012;16:256-65.
- 127. Rapues J, Wilson EC, Packer T, Colfax GN, Raymond HF. Correlates of HIV infection among transfemales, San Francisco, 2010: results from a respondent-driven sampling study. Am J Public Health 2013;103:1485-92.


- 128. Santos GM, Das M, Santos D, Chu P, Colfax G. Social network analysis of methamphetamine-using men who have sex with men in San Francisco. 2011 National HIV Prevention Conference Abstract# 1463 Atlanta, GA2011.
- 129. Santos GM, Rapues J, Wilson EC, et al. Alcohol and substance use among transgender women in San Francisco: Prevalence and association with human immunodeficiency virus infection. Drug Alcohol Rev 2014.
- 130. Santos GM, Do T, Beck J, et al. Syndemic conditions associated with increased HIV risk in a global sample of men who have sex with men. Sex Transm Infect 2014;90:250-3.
- 131. Santos GM, Beck J, Wilson PA, et al. Homophobia as a barrier to HIV prevention service access for young men who have sex with men. J Acquir Immune Defic Syndr 2013;63:e167-70.
- 132. Johnston LG, Prybylski D, Raymond HF, Mirzazadeh A, Manopaiboon C, McFarland W. Incorporating the service multiplier method in respondent-driven sampling surveys to estimate the size of hidden and hard-to-reach populations: case studies from around the world. Sex Transm Dis 2013;40:304-10.
- 133. Silva-Santisteban A, Raymond HF, Salazar X, et al. Understanding the HIV/AIDS epidemic in transgender women of Lima, Peru: results from a sero-epidemiologic study using respondent driven sampling. AIDS Behav 2012;16:872-81.
- 134. Malekinejad M, McFarland W, Vaudrey J, Raymond HF. Accessing a diverse sample of injection drug users in San Francisco through respondent-driven sampling. Drug Alcohol Depend 2011;118:83-91.
- 135. Kral AH, Malekinejad M, Vaudrey J, et al. Comparing respondent-driven sampling and targeted sampling methods of recruiting injection drug users in San Francisco. J Urban Health 2010;87:839-50.
- 136. Ma X, Zhang Q, He X, et al. Trends in prevalence of HIV, syphilis, hepatitis C, hepatitis B, and sexual risk behavior among men who have sex with men. Results of 3 consecutive respondent-driven sampling surveys in Beijing, 2004 through 2006. J Acquir Immune Defic Syndr 2007;45:581-7.
- 137. Wei C, McFarland W, Colfax GN, Fuqua V, Raymond HF. Reaching black men who have sex with men: a comparison between respondent-driven sampling and time-location sampling. Sex Transm Infect 2012;88:622-6.
- 138. Harris DS, Batki SL, Berger SP. Fluoxetine attenuates adrenocortical but not subjective responses to cocaine cues. Am J Drug Alcohol Abuse 2004;30:765-82.
- 139. Batki SL, Washburn AM, Delucchi K, Jones RT. A controlled trial of fluoxetine in crack cocaine dependence. Drug Alcohol Depend 1996;41:137-42.
- 140. Batki SL, Manfredi LB, Jacob P, 3rd, Jones RT. Fluoxetine for cocaine dependence in methadone maintenance: quantitative plasma and urine cocaine/benzoylecgonine concentrations. J Clin Psychopharmacol 1993;13:243-50.
- 141. Batki SL. Review: antidepressants are not effective for cocaine dependence. Evid Based Ment Health 2002;5:82-3.
- 142. Batki SL. Review: dopamine agonists are not effective for cocaine dependence. Evid Based Ment Health 2002;5:82-3.
- 143. Latkin CA, Mandell W, Vlahov D. The relationship between risk networks' patterns of crack cocaine and alcohol consumption and HIV-related sexual behaviors among adult injection drug users: a prospective study. Drug Alcohol Depend 1996;42:175-81.
- 144. Factor SH, Wu Y, Monserrate J, et al. Drug use frequency among street-recruited heroin and cocaine users in Harlem and the Bronx before and after September 11, 2001. J Urban Health 2002;79:404-8.
- 145. Coffin PO, Galea S, Ahern J, Leon AC, Vlahov D, Tardiff K. Opiates, cocaine and alcohol combinations in accidental drug overdose deaths in New York City, 1990-98. Addiction 2003;98:739-47.


- 146. Fuller CM, Absalon J, Ompad DC, et al. A comparison of HIV seropositive and seronegative young adult heroin- and cocaine-using men who have sex with men in New York City, 2000-2003. J Urban Health 2005;82:i51-61.
- 147. Lai S, Lima JA, Lai H, et al. Human immunodeficiency virus 1 infection, cocaine, and coronary calcification. Arch Intern Med 2005;165:690-5.
- 148. Galea S, Nandi A, Coffin PO, et al. Heroin and cocaine dependence and the risk of accidental non-fatal drug overdose. J Addict Dis 2006;25:79-87.
- 149. Amesty S, Ompad DC, Galea S, et al. Prevalence and correlates of previous hepatitis B vaccination and infection among young drug-users in New York City. J Community Health 2008;33:139-48.
- 150. Colfax G, Santos GM, Chu P, et al. Amphetamine-group substances and HIV. Lancet 2010;376:458-74.
- 151. Heckathorn DD. Extensions of responder-driven sampling: analyzing continuous variables and controlling for differential recruitment. Sociol Methodol 2007;37:151-207.
- 152. Magnani R, Sabin K, Saidel T, Heckathorn D. Review of sampling hard-to-reach and hidden populations for HIV surveillance. AIDS 2005;19 Suppl 2:S67-72.
- 153. Wejnert C, Heckathorn DD. Web-Based Network Sampling. Sociological Methods & Research 2008;37:105-34.
- 154. McKnight C, Des Jarlais D, Bramson H, et al. Respondent-driven sampling in a study of drug users in New York City: notes from the field. J Urban Health 2006;83:i54-9.
- 155. McCann DJ, Petry NM, Bresell A, Isacsson E, Wilson E, Alexander RC. Medication Nonadherence, "Professional Subjects," and Apparent Placebo Responders: Overlapping Challenges for Medications Development. J Clin Psychopharmacol 2015;35:566-73.
- 156. Devine EG, Waters ME, Putnam M, et al. Concealment and fabrication by experienced research subjects. Clinical trials 2013;10:935-48.
- 157. Smith SR, Prosser WA, Donahue DJ, et al. Lorcaserin (APD356), a selective 5-HT(2C) agonist, reduces body weight in obese men and women. Obesity (Silver Spring) 2009;17:494-503.
- 158. Fals-Stewart W, O'Farrell TJ, Freitas TT, McFarlin SK, Rutigliano P. The timeline followback reports of psychoactive substance use by drug-abusing patients: psychometric properties. J Consult Clin Psychol 2000;68:134-44.
- 159. Kranzler HR, Tennen H, Armeli S, et al. Targeted naltrexone for problem drinkers. J Clin Psychopharmacol 2009;29:350-7.
- 160. Haberer JE, Kahane J, Kigozi I, et al. Real-time adherence monitoring for HIV antiretroviral therapy. AIDS Behav 2010;14:1340-6.
- 161. Turner C, Coffin PO, Santos DM, et al. Race/ethnicity and education predict engagement in text messaging: Digital divide in ecological momentary assessments among substance-using MSM in San Francisco. In: Francisco UoCS, ed. University of California San Francisco Health Disparities Research Symposium IX. San Francisco, CA2015.
- 162. Preston KL, Silverman K, Schuster CR, Cone EJ. Assessment of cocaine use with quantitative urinalysis and estimation of new uses. Addiction 1997;92:717-27.
- 163. Kiluk BD, Carroll KM, Duhig A, et al. Measures of outcome for stimulant trials: ACTTION recommendations and research agenda. Drug Alcohol Depend 2016;158:1-7.
- 164. Spiehler V, Fay J, Fogerson R, Schoendorfer D, Niedbala RS. Enzyme immunoassay validation for qualitative detection of cocaine in sweat. Clinical chemistry 1996;42:34-8.
- 165. Preston KL, Huestis MA, Wong CJ, Umbricht A, Goldberger BA, Cone EJ. Monitoring cocaine use in substance-abuse-treatment patients by sweat and urine testing. Journal of analytical toxicology 1999;23:313-22.
- 166. Kamb ML, Fishbein M, Douglas JM, Jr., et al. Efficacy of risk-reduction counseling to prevent human immunodeficiency virus and sexually transmitted diseases: a randomized controlled trial. Project RESPECT Study Group. Jama 1998;280:1161-7.


- 167. Brief D, Bollinger, A., Horton, G. & LoCastro, J. S. Relapse Prevention Treatment for Cocaine Addiction: the RPT-C Manual. Bethesda, MD: Medication Development Division, National Institute on Drug Abuse; 1998.
- 168. Miller W, Rollnick S. Motivational Interviewing. 2nd ed. New York: Guilford Press; 2002.
- 169. Miller WR. Motivational interviewing with problem drinkers. Behavioural Psychotherapy 1983;11:147-72.
- 170. DiClemente CC, Prochaska JO, Gilbertini M. Self-efficacy and the stages of self change in smoking. Cognitive Therapy and Research 1985;9:181-200.
- 171. Dunn C, Deroo L, Rivara FP. The use of brief interventions adapted from motivational interviewing across behavioral domains: a systematic review. Addiction 2001;96:1725-42.
- 172. Samet JH, Rollnick S, Barnes H. Beyond CAGE. A brief clinical approach after detection of substance abuse. Arch Intern Med 1996;156:2287-93.
- 173. Rollnick S, Miller W. What is motivational interviewing? Cognit Behav Psychother 1995;25:325-34.
- 174. Kampman KM, Leiderman D, Holmes T, et al. Cocaine Rapid Efficacy Screening Trials (CREST): lessons learned. Addiction 2005;100:102-10.
- 175. Shoptaw S, Reback CJ, Peck JA, et al. Behavioral treatment approaches for methamphetamine dependence and HIV-related sexual risk behaviors among urban gay and bisexual men. Drug and Alcohol Dependence 2005;78:125-34.
- 176. Rawson RA, Marinelli-Casey P, Anglin MD, et al. A multi-site comparison of psychosocial approaches for the treatment of methamphetamine dependence. Addiction 2004;99:708-17.
- 177. U.S. Department of Health and Human Services NIoH, National Institute of Allergy and Infectious Diseases, Division of AIDS, . Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0. 2014.
- 178. Koblin B, Chesney M, Coates T, et al. Effects of a behavioural intervention to reduce acquisition of HIV infection among men who have sex with men: the EXPLORE randomised controlled study. Lancet 2004;364:41-50.
- 179. Macalino GE, Celentano DD, Latkin C, Strathdee SA, Vlahov D. Risk behaviors by audio computer-assisted self-interviews among HIV-seropositive and HIV-seronegative injection drug users. AIDS Educ Prev 2002;14:367-78.
- 180. Hunt MK, Hopko DR, Bare R, Lejuez CW, Robinson EV. Construct validity of the Balloon Analog Risk Task (BART): associations with psychopathy and impulsivity. Assessment 2005;12:416-28.
- 181. Wingrove J, Bond AJ. Impulsivity: A State as Well as Trait Variable. Does Mood Awareness Explain Low Correlations Between Trait and Behavioral Measures of Impulsivity. Person Individ Diff 1997;22:333-9.
- 182. Bancroft J, Vukadinovic Z. Sexual addiction, sexual compulsivity, sexual impulsivity, or what? Toward a theoretical model. J Sex Res 2004;41:225-34.
- 183. Cheng ST, Chan AC, Fung HH. Factorial structure of a short version of the Center for Epidemiologic Studies Depression Scale. Int J Geriatr Psychiatry 2006;21:333-6.
- 184. Gossop M, Darke S, Griffiths P, et al. The Severity of Dependence Scale (SDS): psychometric properties of the SDS in English and Australian samples of heroin, cocaine and amphetamine users. Addiction 1995;90:607-14.
- 185. Tziortzis D, Mahoney JJ, 3rd, Kalechstein AD, Newton TF, De La Garza R, 2nd. The relationship between impulsivity and craving in cocaine- and methamphetamine-dependent volunteers. Pharmacol Biochem Behav 2011;98:196-202.
- 186. Halikas JA, Kuhn KL, Crosby R, Carlson G, Crea F. The measurement of craving in cocaine patients using the Minnesota Cocaine Craving Scale. Comprehensive psychiatry 1991;32:22-7.
- 187. Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med 2001;33:337-43.


- 188. Charmaz K. Premises, principles, and practices in qualitative research: revisiting the foundations. Qual Health Res 2004:14:976-93.
- 189. Strauss AL. Qualitative analysis for social scientists. Cambridge: Cambridge University Press; 1987.
- 190. Morse JM, Barrett M, Mayan M, Olson K, Spiers J. Verification strategies for establishing reliability and validity in qualitative research. International Journal of Qualitative Methods 2002;1:1-19.
- 191. Denzin NK, Lincoln YS. Strategies of qualitative inquiry: Sage; 1998.
- 192. Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol 2004;159:702-6.
- 193. Cole SR, Hernan MA. Fallibility in estimating direct effects. Int J Epidemiol 2002;31:163-5.
- 194. Robins JM, Hernan MA, Brumback B. Marginal structural models and causal inference in epidemiology. Epidemiology 2000;11:550-60.
- 195. Hernan MA, Brumback B, Robins JM. Marginal structural models to estimate the joint causal effect of nonrandomized treatments. J Amer Stat Assoc 2001;96:440-8.
- 196. McCann DJ, Li SH. A Novel, Nonbinary Evaluation of Success and Failure Reveals Bupropion Efficacy Versus Methamphetamine Dependence: Reanalysis of a Multisite Trial. CNS Neurosci Ther 2011.
- 197. Schedules of Controlled Substances: Placement of Lorcaserin Into Schedule IV. Drug Enforcement Administration, 2013. (Accessed December 22, 2014, 2014, at <a href="https://www.federalregister.gov/articles/2013/05/08/2013-10895/schedules-of-controlled-substances-placement-of-lorcaserin-into-schedule-iv">https://www.federalregister.gov/articles/2013/05/08/2013-10895/schedules-of-controlled-substances-placement-of-lorcaserin-into-schedule-iv</a>.)
- 198. Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry 2006;63:484-9.
- 199. Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. Journal of psychiatric research 2011;45:626-9.
- 200. National Institute on Drug Abuse. 2016-2020 NIDA Strategic Plan Advancing Addiction Science: Priority Focus Areas. Rockville, Maryland2015 December 1, 2015.
- 201. Halpern B, Halpern A. Safety assessment of FDA-approved (orlistat and lorcaserin) antiobesity medications. Expert opinion on drug safety 2015;14:305-15.
- 202. Frank C. Recognition and treatment of serotonin syndrome. Canadian family physician Medecin de famille canadien 2008;54:988-92.
- 203. Dunkley EJ, Isbister GK, Sibbritt D, Dawson AH, Whyte IM. The Hunter Serotonin Toxicity Criteria: simple and accurate diagnostic decision rules for serotonin toxicity. QJM: monthly journal of the Association of Physicians 2003;96:635-42.
